Official Title: Benefits of a Long Term Implantable Continuous Glucose Monitoring System for Adults with Diabetes France Adoption Randomized Clinical Trial

NCT Number: NCT03445065

**Document Date:** SAP Version 2.0: 30-Sept-2020

| Roche Diabetes Care | Statistical Analysis Plan | Dago 1 / 64 |
|---------------------|---------------------------|---------------------------|
| EVERSENSE | Version 2.0 – 30/09/2020 | Page <b>1</b> / <b>64</b> |

# **EVERSENSE**

# Benefits of a Long Term implantable Continuous Glucose Monitoring System for Adults with Diabetes France Adoption Randomized Clinical Trial

# STATISTICAL ANALYSIS PLAN

Version 2.0 – 30/09/2020 Written by RCTs

# **Table of contents**

| TΑ | BLE OF CON | FENTS | 2 |
|---|---|---|---|
| 1. | STATISTIC | AL ANALYSIS PLAN - APPROVAL FORM | 5 |
| 2. | VERSION | HISTORY | 6 |
| 3. | ABBREVI <i>A</i> | ATIONS | 7 |
| 4. | | )L | |
| 5. | | SETS AND SUBGROUPS | |
| | | YSIS SETS | |
| | | DRT ANALYSED | |
| | 5.3. FOLL | OW-UP GROUP | 9 |
| 6. | ENDPOIN | TS | 10 |
| | - | ARY EFFICACY ENDPOINT | _ |
| | | NDARY EFFICACY ENDPOINTS | |
| | 6.2.1. | Safety of the insertion and removal procedures and safety of the device | |
| | 6.2.2. | Percentage of time spent in the [70mg/dL-180mg/dL] glucose range | |
| | 6.2.3.<br>6.2.4. | Percentage of time spent in hypoglycemia and hyperglycemia | |
| | | to mean daily glucoseto mean daily glucose | |
| | 6.2.4.1. | Coefficient of variation (CV) | |
| | 6.2.4.2. | Blood Glucose Index | |
| | 6.2.5. | Sensor life | |
| | 6.2.6. | Transmitter wear time | |
| | 6.2.7. | Availability of sensor data | 13 |
| | 6.2.8. | Frequency of access of app pages | 13 |
| | 6.2.9. | Frequency and type of alarms/alerts received | 13 |
| | 6.2.10. | HbA1C (%) level | |
| | 6.2.11. | Maintain of the Eversense effect on hypoglycemia between D150 and D180 for enabled gro<br>15 | · |
| | 6.2.12. | Comparison of data from D90-D120 period to D150-D180 period for control group | |
| | 6.2.13. | Patient Reported Outcome Measures (PROMs) | |
| | 6.2.13.1<br>6.2.13.2 | • | |
| | 6.2.13.2 | | |
| | 6.2.13.4 | | |
| | 6.2.13.5 | · | |
| | 6.2.13.6 | 71 07 | |
| | 6.2.13.7 | | |
| | 6.2.13.8 | . Free text questionnaire for 'enabled' patients only to record the opinion of the patient about the<br>d' system | |
| | 6.2.13.9 | • | |
| | | ators about the system | |
| | 6.3. SAFE | TY ENDPOINTS | 19 |
| | 6.3.1. | Adverse events | 19 |
| | 6.4. Отн | R ENDPOINTS AND VARIABLES | |
| | 6.4.1. | Demographic data and other baseline characteristics | |
| | 6.4.2. | Follow-up data | |
| | 6.4.3. | Medical history | |
| | 6.4.4. | Prior and concomitant therapies | |
| | 6.4.5. | Extent of exposure | |
| 7. | DATA AN | ALYSIS CONSIDERATIONS | 24 |

| 7 | 7.1. ST | ATISTICAL SOFTWARE | 24 |
|---|---|---|---|
| - | 7.2. Ty | PE I ERROR, HANDLING OF MULTIPLICITY ISSUES AND ALPHA ADJUSTMENT PROCEDURES | 24 |
| 7 | 7.3. CE | NTER EFFECT AND POOLING OF CENTERS | 24 |
| - | 7.4. DE | SCRIPTIVE ANALYSES OF QUANTITATIVE AND QUALITATIVE VARIABLES | 24 |
| - | 7.5. DE | FINITION OF BASELINE, TIME-WINDOWS AND ANALYSIS PERIODS | 25 |
| - | 7.6. H <i>i</i> | ANDLING OF MISSING DATA AND INTERCURRENT EVENTS | 26 |
| 8. | | ED STATISTICAL ANALYSES | |
| | | SPOSITION OF PATIENTS | |
| | - | OTOCOL DEVIATIONS | |
| | - | IALYSIS SETS AND COHORTS ANALYZED. | |
| | | MOGRAPHIC DATA AND BASELINE CHARACTERISTICS, INCLUDING MEDICAL HISTORY AND THERAPIES | |
| • | 8.4.1. | Analysis of demographic data and other baseline characteristics | |
| | 8.4.2. | Analysis of follow-up data | |
| | 8.4.3. | Analysis of Medical and surgical history | |
| | 8.4.4. | Analysis of Prior and concomitant therapies | |
| , | _ | IALYSIS OF EXTENT OF EXPOSURE AND TREATMENT COMPLIANCE | |
| Č | | FICACY ANALYSIS | |
| | 8.6.1. | Analysis of the primary efficacy endpoint | |
| | 8.6.1.<br>8.6.1. | | |
| | 8.6.2. | Analysis of the secondary efficacy endpoints | |
| | 8.6.2. | | |
| | 8.6.2. | | |
| | 8.6.2. | | |
| | 8.6.2. | | |
| | stand | ard deviation to mean daily glucose | 42 |
| | 8.6 | 5.2.4.1. Analysis of Coefficient of Variation | 42 |
| | | 5.2.4.2. Analysis of Blood Glucose Indexes | |
| | 8.6.2. | , | |
| | 8.6.2. | , | |
| | 8.6.2. | | |
| | 8.6.2. | , | |
| | 8.6.2.<br>8.6.2. | | |
| | 8.6.2. | · | |
| | 8.6.2. | | |
| | 8.6.2. | | |
| | 8.6.2. | | |
| 8 | 8.7. SA | FETY ANALYSIS | |
| | 8.7.1. | Adverse events | |
| | 8.7.1. | 1. Overall summary of adverse events | 51 |
| | 8.7.1. | 2. Analysis of adverse events by MedDRA coding | 52 |
| | 8.7.1. | 3. Analysis of adverse events per 100 patient years | 53 |
| 8 | 8.8. Ini | DIVIDUAL DATA LISTINGS | 55 |
| | 8.8.1. | Disposition of patients – all patients | 55 |
| | 8.8.2. | Protocol deviations – all patients | 55 |
| | 8.8.3. | Analysis sets and cohorts analyzed – all patients | 56 |
| | 8.8.4. | Demographic data and other baseline characteristics, including medical history and therapies | s — |
| | all patie | nts | 56 |
| | 8.8.5. | Extent of exposure and treatment compliance | 57 |
| | 8.8.6. | Primary efficacy endpoint | |
| | 8.8.6. | | |
| | 8.8.6. | 7,10,711 | |
| | 8.8.7. | Secondary efficacy endpoint | |
| | 8.8.8. | Adverse events | 58 |
| 9. | ДІ СОРІ | THMS | 50 |
| J. | YFOOVI | I I II II I I I I I I I I I I I I I I | |

| Roche Diabetes Care | Statistical Analysis Plan | Daga 4 / 64 |
|---------------------|---------------------------|--------------------|
| EVERSENSE | Version 2.0 – 30/09/2020 | Page <b>4 / 64</b> |

| 9.1. | HANDLING OF MISSING CGM DATA | 59 |
|---|---|---|
| 9.2. | COMPUTATION RULES FOR TIME SPENT IN-, BELOW- AND ABOVE- TARGET RANGES | 60 |
| 10. | CHANGES IN THE STATISTICAL METHODS FROM THOSE STATED IN THE PROTOCOL | 62 |
| 11. | QUALITY CONTROL | 63 |
| 12. | REFERENCES | 64 |

| Roche Diabetes Care | Statistical Analysis Plan | Page 5 / 64 |
|---------------------|---------------------------|-------------|

# 1. STATISTICAL ANALYSIS PLAN - APPROVAL FORM



| Function | Name | Signature | Date |
|----------|------|---------------------------|--------------|
| | | Sep 30, 2020 08:56 GMT+2) | Sep 30, 2020 |

# Scientific committee

| Function | Name | Signature | Date |
|------------------------|-------|-----------|-------------|
| Principal investigator | Prof. | | |
| | | | Oct 1, 2020 |



| Function | Name | Signature | Date |
|----------|------|-----------|-------------|
| | | | Oct 7, 2020 |

| Roche Diabetes Care | Statistical Analysis Plan | Dago 6 / 64 |
|---------------------|---------------------------|--------------------|
| EVERSENSE | Version 2.0 – 30/09/2020 | Page <b>6 / 64</b> |

# 2. VERSION HISTORY

| Version | Date | Author | Comment / changes |
|---|---|---|---|
| 0.1 | 30/04/2019 | RCTs | Initial draft version (based on protocol v5.0 dated of 11/12/2018) |
| 0.2 | 03/07/2019 | RCTs | Including comments from Roche Diabetes Care (France) |
| 0.3 | 09/10/2019 | RCTs | Including comments from Roche Diabetes Care (France) |
| 0.4 | 29/11/2019 | RCTs | Including lasts comments from Roche Diabetes Care (France) |
| 0.5 | 13/12/2019 | RCTs | Including comments from Roche Diabetes Care (France) |
| 1.0 | 28/01/2020 | RCTs | Final version |
| 1.1 | 29/09/2020 | RCTs | Revised version following Data Review meeting |
| 2.0 | 30/09/2020 | RCTs | Final version 2.0 |

| Roche Diabetes Care | Statistical Analysis Plan | Daga 7 / 64 |
|---------------------|---------------------------|--------------------|
| EVERSENSE | Version 2.0 – 30/09/2020 | Page <b>7 / 64</b> |

# 3. ABBREVIATIONS

| Abbreviation | Description |
|--------------|----------------------------------------------------|
| ADDQoL | Audit of Diabetes Dependent Quality of Life |
| ADE | Adverse device effect |
| AE | Adverse event |
| ATC | Anatomical Therapeutic Chemical |
| BG | Blood Glucose |
| BGRI | Blood Glucose Risk Index |
| BOCF | Baseline Observation Carried Forward |
| CGM-Sat | Continuous Glucose Monitoring – Satisfaction scale |
| CI | Confidence interval |
| CV | Coefficient of Variation |
| eCRF | Electronic case report form |
| FAS | Full analysis set |
| FGM | Flash glucose monitoring |
| GLM | Generalized Linear Model |
| HbA1c | Glycated hemoglobin |
| HBGI | High Blood Glucose Index |
| INN | International nonproprietary name |
| IRB | Independent review board |
| ITT | Intent-to-treat |
| LBGI | Low Blood Glucose Index |
| LLN | Lower limit of normal |
| LLT | Lowest level term |
| LOCF | Last observation carried forward |
| MedDRA | Medical Dictionary for Regulatory Activities |
| CGM | Continuous glucose monitoring |
| MNAR | Missing not at random |
| MD | Missing data |
| MDP | Missing data pattern |
| PP | Per protocol |
| PT | Preferred term |

| Roche Diabetes Care | Statistical Analysis Plan | Daga 9 / 64 |
|---------------------|---------------------------|--------------------|
| EVERSENSE | Version 2.0 – 30/09/2020 | Page <b>8 / 64</b> |

| Abbreviation | Description |
|--------------|-------------------------------------------|
| Q1 | First quartile |
| Q3 | Third quartile |
| SAE | Serious adverse event |
| SAP | Statistical analysis plan |
| SD | Standard deviation |
| SOC | System organ class |
| TEAE | Treatment emerged adverse events |
| UADE | Unanticipated Adverse Device Effect |
| WHO-DD | World Health Organization drug dictionary |

| Roche Diabetes Care | Statistical Analysis Plan | Daga 0 / 64 |
|---------------------|---------------------------|--------------------|
| EVERSENSE | Version 2.0 – 30/09/2020 | Page <b>9 / 64</b> |

# 4. PROTOCOL

This Statistical Analysis Plan refers to protocol version 5.0 dated December 11th, 2018.

# 5. ANALYSIS SETS AND SUBGROUPS

# 5.1. Analysis sets

The analysis sets are defined below:

- **Screened Set:** The Screened Set population consists of all patients who signed an informed consent.
- Randomized Set (RS): The Randomized Set consists of all patients from the Screened Set who
  have been randomized.
- Full Analysis Set (FAS): The FAS population consists of all randomized patients with the sensor inserted at Visit 2 (D0) and with at least one CGM data available from randomization visit to D180 visit. This is the primary population for the analysis of efficacy.
- **Per-Protocol (PP):** The Per-Protocol population consists of all FAS patients without major protocol deviation, defined blindly by the scientific committee during the data review before the data base lock (see Section 8.2 for definition of major protocol deviations).
- Safety Set (SAF): The Safety Set consists of all patients with the sensor inserted at Visit 2 (D0). This is the primary population for the analysis of safety.

# 5.2. Cohort analysed

The following cohorts are defined according to the type of diabetes or HbA1c (%) level during selection phase and will be studied:

- **Cohort 1:** patients with HbA1c level > 8.0% (either type 1 or type 2 diabetes)
- **Cohort 2:** patients having type 1 diabetes and spending more than 1.5 hour with FGM <70 mg/dl per day as a mean for at least 28 days.

# 5.3. Follow-up group

According to protocol section 2.1, patients selected in cohort 2 at D0 who no longer comply with the inclusion criteria (i.e. spend more than 1.5 hour with FGM <70 mg/dl per day as a mean for at least 28 days) at D30, will have the opportunity to start using the system, but in an open phase, the investigator will determine the planning of visits as per their usual follow-up, no data will be collected except the report of any adverse event.

The follow-up group will be computed as follows:

- Patients pre-selected in cohort 2 at D0 (i.e. Type 1 Diabetes and spend more than 1.5 hour with FGM <70 mg/dl per day as a mean for at least 28 days), and</li>
- Patients not randomized, and
- Patients with date of end of study (\*) > date of D30.

(\*) with date of end of study defined as the minimum between date of study withdrawal, consent withdrawal, last contact date, or death.

| Roche Diabetes Care | Statistical Analysis Plan | Daga 10 / 64 |
|---------------------|---------------------------|---------------------|
| EVERSENSE | Version 2.0 – 30/09/2020 | Page <b>10 / 64</b> |

# 6. ENDPOINTS

Unless otherwise specified, endpoints will be computed per patient (i.e. the statistical unit is the patient).

# 6.1. Primary efficacy endpoint

As described in protocol section 14.4, "the primary efficacy objective for **cohort 1** is to evaluate the difference between Enabled and Control arms in HbA1c (%) level at D180". Analysis of the primary endpoint for Cohort 1 is described in Section 8.6.1.1.

For **cohort 2**, the primary efficacy objective is to evaluate the difference between Enabled and Control arms in percentage of time spent in hypoglycemia < 54 mg/dl between D90 visit and D120 visit (using CGM system data). Analysis of the primary endpoint for Cohort 2 is described in Section 8.6.1.2.

This endpoint will be computed as follows:

Percentage of time spent in hypoglycemia < 54mg/dL =</li>

```
100* \frac{duration (min) spent with glycemia < 54 mg/dL between D90 and D120}{duration (min) with CGM data available (i.e. excluding temporary discontinuations)}
```

The algorithm is defined in section 9.2.

# 6.2. Secondary efficacy endpoints

Unless otherwise specified, the following secondary efficacy criteria will be computed for both cohorts.

# 6.2.1. Safety of the insertion and removal procedures and safety of the device

The following pre-specified AE reported in the eCRF from D0 to D187 will be used:

- Infection, local or systemic
- Excessive bleeding
- Bruising or swelling
- Keloid and/or scar formation
- Skin irritation and/or redness
- Nerve damage causing tingling, numbness, pain or weakness
- Puritis (itching of the incision while healing)
- Discoloration of skin
- Hematoma formation
- Burning sensation or pain
- Device migration

Pre-specified AE which occurred after sensor insertion and after sensor removal will be analyzed separately.

# 6.2.2. Percentage of time spent in the [70mg/dL-180mg/dL] glucose range

From D90 to D120

| Roche Diabetes Care | Statistical Analysis Plan | Page 11 / 64 |
|---------------------|---------------------------|---------------------|
| EVERSENSE | Version 2.0 – 30/09/2020 | Page <b>11 / 64</b> |

From D150 to D180

These endpoints will be computed using CGM data. The algorithm is defined in section 9.2.

See Section 7.5 for definition of time-windows D90-D120 and D150-D180.

# 6.2.3. Percentage of time spent in hypoglycemia and hyperglycemia

The following endpoints will be computed using CGM data. The algorithm is defined in section 9.2.

- Hypoglycemia (<70mg/dL) from D90 to D120</li>
- Hypoglycemia (<70mg/dL) from D150 to D180</li>
- Hypoglycemia (<54mg/dL) from D90 to D120</li>
- Hypoglycemia (<54mg/dL) from D150 to D180</li>
- Hyperglycemia (>180mg/dL) from D90 to D120
- Hyperglycemia (>180mg/dL) from D150 to D180
- Hyperglycemia (>250mg/dL) from D90 to D120
- Hyperglycemia (>250mg/dL) from D150 to D180

See Section 7.5 for definition of time-windows D90-D120 and D150-D180.

# 6.2.4. Glucose variability estimated with coefficient of variation calculated by 24h as ratio of standard deviation to mean daily glucose

Glucose variability will be evaluated using the following indices.

#### 6.2.4.1. Coefficient of variation (CV)

#### CV measured from D90 to D120:

This endpoint will be computed using CGM data with the following formula.

$$Coefficient \ of \ variation \ (\%) = \frac{\sum_{i=90}^{i=120} \frac{SD_i}{Mean_i}}{n} * 100$$

# Where

- SD<sub>i</sub> = Standard deviation of CGM glycemia measured values on Day i,
- Mean<sub>i</sub> = mean of CGM glycemia measured on Day i,
- Day i starts at 00:00 and stop at 23:59,
- N is the number of days with available CV value.

# CV measured from D90 to D120 will also be classified as ≤36% and >36%:

<u>Note:</u> According to Monnier et al. (1), a CV threshold set to 36% allows to distinguish between stable and unstable glycemia.

#### CV measured from D150 to D180:

Same computation rule.

#### CV measured from D150 to D180 will also be classified as ≤36% and >36%.

| Roche Diabetes Care | Statistical Analysis Plan | Dago 12 / 64 |
|---------------------|---------------------------|---------------------|
| EVERSENSE | Version 2.0 – 30/09/2020 | Page <b>12 / 64</b> |

#### 6.2.4.2. Blood Glucose Index

#### Measured from D90 to D120:

$$LBGI = \frac{1}{N} \sum_{i=1}^{N} rl(BG_i) \qquad HBGI = \frac{1}{N} \sum_{i=1}^{N} rh(BG_i)$$

BGRI = LGBI + HGBI

#### Where:

- BG = Blood Glucose (mg/dL) recorded by the CGM
- BG<sup>new</sup> = 1.509 · ([log(BG)]<sup>1.084</sup> 5.381)
- r(BG) = 10 · BG<sup>new 2</sup>
- rl(BG) = r(BG) if BG<sup>new</sup> < 0 and 0 otherwise</li>
- rh(BG) = r(BG) if BG<sup>new</sup> > 0 and 0 otherwise

Low Blood Glucose Index (LBGI), High Blood Glucose Index (HBGI) and Blood Glucose Risk Index (BGRI) formulas are described by Fabris et Al. (2)

# Measured from D150 to D180:

Same computation rule.

Note: See Section 7.5 for definition of time-windows D90-D120 and D150-D180.

#### 6.2.5. Sensor life

Sensor life will be computed as the number of subjects/Sensors operating at 150- and 180-days post insertion and mean/median Sensor life using Sensor output and long-term performance.

The following endpoints will be computed using CGM data.

- For the first sensor:
  - Lifespan (days) for the first sensor = Date of the last glucose measurement by the sensor – date of the first glucose measurement by the sensor + 1
  - Patients having first sensor operating at D150 (= Yes if lifespan of the first sensor ≥ 150 days, = No otherwise)
  - Patients having first sensor operating at D180 (= Yes if lifespan of the first sensor ≥ 180 days, = No otherwise)
- Number of sensors used (0, 1, 2, 3, etc.)
  - o Between D0 and D180
  - Between D30 and D120
  - o Between D30 and D180

See Section 7.5 for definition of time-windows D0-D180, D30-D120 and D30-D180.

#### 6.2.6. Transmitter wear time

Amount and variability of Transmitter wear time (by day/week/months) will be computed using CGM data.

- For the first transmitter:
  - Lifespan (days) for the first transmitter = Date of the last glucose measurement with the transmitter – date of the first glucose measurement with the transmitter + 1
- Number of transmitters per patients (0, 1, 2, 3, etc.)

| Roche Diabetes Care | Statistical Analysis Plan | Page 12 / 64 |
|---------------------|---------------------------|--------------|

- Between D0 and D180 (or last visit)
- o Between D30 and D120
- Between D30 and D180 (or last visit)

# 6.2.7. Availability of sensor data

This endpoint will be computed for the following studied periods:

- Between D0 and D180
- Between D30 and D120
- Between D30 and D180
- Between D0 and D30
- Between D30 and D60
- Between D60 and D90
- Between D90 and D120
- Between D120 and D150
- Between D150 and D180

Availability of sensor data (%) = 
$$100 * \frac{Duration (min) of available CGM data}{Duration (min) of studied period}$$

If duration of the studied period is missing (i.e. the patient withdrew the study prior to the studied period), the availability of sensor data will be set to missing.

If duration of the studied period is not missing and duration of available CGM data is 0 min (i.e. no CGM data available for the studied period), the availability of sensor data will be set to 0%.

See Section 7.5 for definition of time-windows.

Data downloaded from the CGM file will be used for this purpose.

# 6.2.8. Frequency of access of app pages

This endpoint is not available in CGM files and cannot be computed.

A descriptive analysis of the following data collected in eCRF will be performed:

- Does the patient use the "report" function?
- Does the patient use the "historic of alerts" function?
- Does the patient use the "log event" function?
- · Does the patient use his phone to look at his glucose level?

# 6.2.9. Frequency and type of alarms/alerts received

As patients in cohort 2 will use the CGM in blinded mode, result of this endpoint will be provided for cohort 1 only.

Measured from D0 to D187: this endpoint is defined as the number of alarms received by the patient (for each type of alarm and overall). This endpoint will be computed using data downloaded from the CGM system. The type of alarms recorded in CGM system are the following:

| Roche Diabetes Care | Statistical Analysis Plan | Dogo 14 / 64 |
|---------------------|---------------------------|--------------|

| Group | Alarm type | Message | Received alert |
|---|---|---|---|
| READER<br>ERROR | Sensor related | Ambient Light Warning | High Ambient Light Alert |
| | Calibration | Calibration Expired Alarm<br>Asserted | Calibration Expired |
| | Calibration | Calibration Grace Period Alarm<br>Asserted | Calibration Past Due |
| | Sensor Glucose | Falling Rate Alert Asserted | Rate Falling |
| | Sensor Glucose | High Glucose Alarm Asserted | Hight Glucose |
| READER | Sensor Glucose | Invalid High Glucose Asserted | Out of Range High Glucose |
| ALARM | Sensor Glucose | Invalid Low Glucose Asserted | Out of Range Low Glucose |
| | Sensor Glucose | Low Glucose Alarm Asserted | Low glucose |
| | Sensor Glucose | Predictive Falling Rate Alert<br>Asserted | Predicted Low Glucose |
| | Sensor Glucose | Predictive Rising Rate Alert<br>Asserted | Predicted High Glucose |
| | Sensor Glucose | Rising Rate Alert Asserted | Rate Rising |
| | Transmitter related | BLE disconnect event | Transmitter Disconnect |
| | Transmitter related | Critical Fault | Transmitter Error |
| | Transmitter related | High Transmitter Temperature | High Transmitter Temperature |
| READER<br>MISC | System Related | Calibration Phase | Displayed on the Status Bar of the App |
| | Sensor related | High Sensor Temperature | High Sensor Temperature |
| | Sensor related | Low Sensor Temperature | Low Sensor Temperature |
| | Sensor related | MEP Alarm | Sensor Replacement |
| | Sensor related | Sensor Retired | Sensor Replacement |
| | Sensor Glucose and<br>Calibration | Sensor Stability Alarm Activated | Sensor Check |

<u>Note:</u> only messages displayed to the patient are listed in this table. Internal messages (i.e. for engineering use only and not displayed to the patient) are not listed in this table and will not be analyzed.

| Roche Diabetes Care | Statistical Analysis Plan | Dogo 15 / 64 |
|---------------------|---------------------------|---------------------|
| EVERSENSE | Version 2.0 – 30/09/2020 | Page <b>15 / 64</b> |

# 6.2.10. HbA1C (%) level

- HbA1c (%) at D120 visit
- HbA1c (%) at D180 visit for cohort 2 only (see Section 6.1 Primary endpoint for cohort 1).
- HbA1c at D120 visit classified as follows: ≤7% / >7%
- HbA1c at D120 visit classified as follows: ≤6.5% / >6.5%
- HbA1c at D180 visit classified as follows: ≤7% / >7%
- HbA1c at D180 visit classified as follows: ≤6.5% / >6.5%

These endpoints will be studied using data as collected in the eCRF.

# 6.2.11. Maintain of the Eversense effect on hypoglycemia between D150 and D180 for enabled group

The percentage of time spent in hypoglycemia < 54 mg/dl between D150 and D180 will be computed as described in section 6.2.3. This endpoint will be analyzed for patients randomized in Enabled arm of cohort 2 only (cf. section 8.6.2.11).

# 6.2.12. Comparison of data from D90-D120 period to D150-D180 period for control group

The percentage of time spent in hypoglycemia < 54 mg/dl between D90-D120 and between D150-D180 will be computed as described in section 6.2.3. This endpoint will be analyzed for patients randomized in Control arm of cohort 2 only (cf. section 8.6.2.12).

# 6.2.13. Patient Reported Outcome Measures (PROMs)

# 6.2.13.1. CGM questionnaire (CGM SAT)

The CGM-SAT is collected on D60 and D180 for enabled patients only.

44 item scale assessing experiences with CGM over previous 6 months. The scale is designed to measure the impact of CGM on Diabetes management and family relationships, plus on satisfaction with emotional, behavioral and cognitive effects of CGM use. Responses are rated on a 5-point scale from 'strongly disagree' to 'strongly agree'.

Overall score corresponds to the mean of the 44 items. In case of missing items, the overall score will be the mean of available items.

The absolute change in overall CGM-SAT score from D60 to D180 will be computed.

The data will be used as collected in the eCRF.

The validation of this questionnaire used in this study is reported by Tubiana-Rufi (2010).

| Roche Diabetes Care | Statistical Analysis Plan | Dogo 16 / 64 |
|---------------------|---------------------------|---------------------|
| EVERSENSE | Version 2.0 – 30/09/2020 | Page <b>16 / 64</b> |

# 6.2.13.2. Diabetes Treatment Satisfaction Questionnaire original status (DTSQs)

The DTSQs is collected at screening visit, D60 and D180. The DTSQs contains eight items scored on 7-point scale (i.e. each item is scored from 0 to 6).

#### **DTSQs: Treatment Satisfaction score:**

The Treatment Satisfaction score is computed by adding the six items 1, 4, 5, 6, 7 and 8. The Treatment Satisfaction score has a minimum of zero and a maximum of 36.

The absolute changes in Treatment Satisfaction score will be computed:

- from D0 to D180
- from D0 to D60.

#### DTSQs: Items 2 and 3:

Items 2 (Perceived Frequency of Hyperglycemia) and 3 (Perceived Frequency of Hypoglycemia) are treated individually in data analysis. The absolute changes for item 2 and item 3 will be computed:

- from D0 to D180
- from D0 to D60.

# DTSQs: Items 1, 4, 5, 6, 7 and 8:

Each items will be be analyzed separately. For each items, the absolute changes 3 will be computed:

- from D0 to D180
- from D0 to D60.

#### DTSQs: Handling of missing scores on the six Treatment Satisfaction items:

In case of missing items, the Treatment Satisfaction score will be computed as follows:

- Step 1: sum the existing items scores
- Step 2: divide this sum by the number of existing items scores
- Step 3: multiply by 6 (the number of items in the subscale)
- Step 4: use this computation to estimate subscale scores, providing the number of missing values does not exceed the number tolerable without unacceptable loss of reliability for the language version in use.

Note: language version in use is French. The number of tolerable missing items is 3.

#### DTSQs: Handling of missing data for item-by-item analysis:

According to the DTSQ user guidelines, it is recommended to treat a missing score as missing for any item-by-item analyses and do not include computed scores in such analyses. Therefore, missing data will not be replaced for item-by-item analyses.

<u>Note</u>: the reliability and factor structure of the eight language versions used in this study are reported by Plowright (2000).

| Roche Diabetes Care | Statistical Analysis Plan | Dog 17 / 64 |
|---------------------|---------------------------|---------------------|
| EVERSENSE | Version 2.0 – 30/09/2020 | Page <b>17 / 64</b> |

# 6.2.13.3. The Diabetes Treatment Satisfaction Questionnaire change version (DTSQc)

The DTSQc is collected at D180. The DTSQc contains eight items scored on 7-point scale (i.e. each item is scored from -3 to +3).

#### **DTSQc: Treatment Satisfaction score:**

The Treatment Satisfaction score is computed by adding the six items 1, 4, 5, 6, 7 and 8. The Treatment Satisfaction score has a minimum of -18 and a maximum of +18.

#### DTSQc: Items 2 and 3:

Items 2 (Perceived Frequency of Hyperglycemia) and 3 (Perceived Frequency of Hypoglycemia) are treated individually in data analysis.

# DTSQc: Items 1, 4, 5, 6, 7 and 8:

Each items will be analyzed separately.

#### DTSQc: Handling of missing scores on the six Treatment Satisfaction items:

In case of missing items, the Treatment Satisfaction score will be computed as follows:

- Step 1: sum the existing items scores
- Step 2: divide this sum by the number of existing items scores
- Step 3: multiply by 6 (the number of items in the subscale)
- Step 4: use this computation to estimate subscale scores, providing the number of missing values does not exceed the number tolerable without unacceptable loss of reliability for the language version in use.

Note: language version in use is French. The number of tolerable missing items is 3.

# DTSQc: Handling of missing data for item-by-item analysis:

According to the DTSQ user guidelines, it is recommended to treat a missing score as missing for any item-by-item analyses and do not include computed scores in such analyses. Therefore, missing data will not be replaced for item-by-item analyses.

<u>Note</u>: the reliability and factor structure of the eight language versions used in this study are reported by Plowright (2000).

#### 6.2.13.4. The Audit of Diabetes-Dependent Quality of Life (ADDQoL)

The ADDQoL is collected at screening visit and D180.

The ADDQoL measures the impact of diabetes and its treatment on 19 specific aspects of life. The ADDQoL has been designed to permit users to indicate whether potentially affected domains of life apply to them and to rate the impact of their diabetes on all applicable aspects of life, together with the perceived importance of each domain for their QoL.

The scale ranges from -3 to +1 for 19 life domains (impact rating) and from 0 to +3 in attributed importance (importance rating). A weighted score for each domain is calculated as a multiplier of impact rating and importance rating (ranging from -9 to +3). Finally, a mean weighted impact score (ADDQOL score) is calculated for the entire scale across all applicable domains.

The absolute change in overall ADDQOL score from screening visit to D180 will be computed.

The validity and reliability of the 19-item ADDQoL are reported by Wee (2006).

| Roche Diabetes Care | Statistical Analysis Plan | Dago 19 / 64 |
|---------------------|---------------------------|---------------------|
| EVERSENSE | Version 2.0 – 30/09/2020 | Page <b>18 / 64</b> |

# 6.2.13.5. Diabetes Distress Scale 2 (DDS2)

The DDS2 is collected at screening visit, D60 and D180.

The DDS2 is a 2-item diabetes distress screening instrument asking respondents to rate on a 6-point scale the degree to which the following items caused distress: (1) feeling overwhelmed by the demands of living with diabetes, and (2) feeling that I am often failing with my diabetes regimen. Its validation has been published by Fischer (2008).

DDS2 score is the mean of the two items. If one item is missing, then no score will be computed.

In addition, the two items will be analyzed separately.

The absolute change in overall DDS2 score will be computed from screening visit to D60 and from screening visit to D180.

# 6.2.13.6. Hypoglycemia Fear Survey part II (HFS II)

The HFS II – worry scale is collected at screening visit, D60 and D180.

HFS II - worry items describe specific concerns that patients may have about their hypoglycemic episodes (e.g., being alone, episodes occurring during sleep, or having an accident). The scale ranges from 0 (never) to 4 (almost always).

HFS score = Sum of all items.

It is not planned to replace missing items. If one item is missing, the HFS score will not be computed.

The absolute change in overall HFS II score will be computed from screening visit to D60 and from screening visit to D180.

This endpoint will be studied using data collected in the eCRF.

The validity and reliability of the scale are reported by Gonder-Frederick (2011).

# 6.2.13.7. Partner reported Outcome Measures (Partner-DDS) to measure the partner-related distress

This questionnaire is collected at screening visit, D60 and D180.

The Partner-DDS is a 21-item self-report scale that highlights four critical dimensions of partner-related distress: "my partner's diabetes management", "how best to help", "diabetes and me", and "hypoglycemia". The scale ranges from 0 (not at all) to 4 (a great deal).

The PARTNER DDS yields a total diabetes distress score plus 4 subscale scores:

- Total DDS Score = Mean of the 21 items
- My partner's diabetes management = Mean of item 3, 4, 10, 12, 14, 15 and 20
- How best to help = Mean of item 2, 6, 7, 11 and 13
- Diabetes and me = Mean of items 5, 8, 9, 16 and 21
- Hypoglycemia = Mean of items 1, 17, 18 and 19.

The absolute change will be computed from screening visit to D60 and from screening visit to D180 for each score.

The data will be used as collected in the eCRF.

The validity and reliability of the scale are reported by Polonsky (2016).

| Roche Diabetes Care | Statistical Analysis Plan | Page 10 / 64 |
|---------------------|---------------------------|---------------------|
| EVERSENSE | Version 2.0 – 30/09/2020 | Page <b>19 / 64</b> |

# 6.2.13.8. Free text questionnaire for 'enabled' patients only to record the opinion of the patient about the 'enabled' system

This questionnaire is collected at D180 and contains six questions that have the aim to record the opinion of the patient about the 'enabled' system at the end of the study. This questionnaire will add the depth of data and context to the quantitative PRO data that is being collected.

The data will be used as collected in the eCRF.

# 6.2.13.9. Free text questionnaire for study investigators to record the opinion of the principal investigator or co-investigators about the system

This questionnaire is collected at D180 and contains seven questions which have the aim to record the opinion of the principal investigator or co-investigators about the system.

The data will be used as collected in the eCRF.

# 6.3. Safety endpoints

#### 6.3.1. Adverse events

The following adverse events will be studied:

- All adverse events (AE)
- Treatment emergent adverse events (TEAE) [1]
- Serious TEAE
- Fatal TEAE
- Related TEAE (i.e. with possible or probable relationship) to the investigational device according investigator)
- TEAE leading to discontinuation of the investigational device (i.e. temporary or definitive discontinuation)
- TEAE by maximum severity:
  - mild TEAE
  - moderate TEAE
  - severe TEAE

[1] TEAE = AEs occurring on or after the start of the sensor insertion at D0 (Visit 2).

The following AEs will also be studied. Their definition is provided hereafter.

- Symptomatic hypoglycemia
- Severe hypoglycemia (SAEs)
- Serious Diabetic Ketoacidosis (SAEs)
- Adverse Device Effect (ADE) (i.e. anticipated and unanticipated) as collected in the eCRF
  - Anticipated ADE are defined as all AEs which were pre-specified in the eCRF (i.e. Bleedings, Discoloration of skin, Edema or swelling, Hematoma formation, Infection ,local or systemic, Itching and / or puritis, Nerve damage causing tingling, numbness, pain or weakness, Pain and / or burning sensation, Skin irritation and / or redness, ...)

| Roche Diabetes Care | Statistical Analysis Plan | Page <b>20</b> / 64 |
|---------------------|---------------------------|---------------------|
| EVERSENSE | Version 2.0 – 30/09/2020 | Page <b>20 / 64</b> |

- Unanticipated ADE are defined as all related AEs (i.e. with possible or probable relationship) which were not pre-specified in the eCRF.
- ADE as reported to the hotline

•

# **Programming definitions:**

Hypoglycemia will be identified in AE forms using the following Standardized MedDRA Queries (SMQ)

| SMQ: Hypoglycaemia<br>SMQ code: 20000226<br>Narrow definition | |
|---------------------------------------------------------------|----------|
| PT | PT code |
| Blood glucose decreased | 10005555 |
| Hyperinsulinaemic hypoglycaemia | 10077216 |
| Hypoglycaemia | 10020993 |
| Hypoglycaemia neonatal | 10020994 |
| Hypoglycaemia unawareness | 10020997 |
| Hypoglycaemic coma | 10021000 |
| Hypoglycaemic encephalopathy | 10021002 |
| Hypoglycaemic seizure | 10048803 |
| Hypoglycaemic unconsciousness | 10065981 |
| Nesidioblastosis | 10080024 |
| Neuroglycopenia | 10054998 |
| Postprandial hypoglycaemia | 10059035 |
| Shock hypoglycaemic | 10040576 |

<u>Symptomatic hypoglycemia</u>: all hypoglycemia reported in AE forms will be considered as symptomatic.

<u>Severe hypoglycemia</u>: all hypoglycemia reported in AE forms with item Serious = Yes and Intensity = "Severe" or "Life threatening".

As define in section 11.2.2 of the protocol, a severe hypoglycemia episode is defined as symptoms in loss of consciousness and/or seizures resolving upon administration of glucose or glucagon by another person (only third-party assistance). It usually requires needing assistance that can require in addition medical attention (emergency room, hospitalization). Severe hypoglycemia are defined as SAEs.

Serious Diabetic Ketoacidosis will be identified in AE forms using the following MedDRA terms:

| Roche Diabetes Care | Statistical Analysis Plan | Dogo 31 / 64 |
|---------------------|---------------------------|---------------------|
| EVERSENSE | Version 2.0 – 30/09/2020 | Page <b>21 / 64</b> |

| System Organ<br>Class<br>(SOC Code) | Preferred Term<br>(PT Code) | Lowest Level Term<br>(LLT Code) |
|---|---|---|
| Metabolism and nutrition | Euglycaemic diabetic ketoacidosis (10080061) | Euglycaemic diabetic ketoacidosis (10080061) Euglycemic diabetic ketoacidosis (10080062) |
| disorders<br>(10027433) | Diabetic ketoacidosis<br>(10012671) | Acidosis diabetic (10000488) Diabetes mellitus with ketoacidosis (10012622) Diabetes with ketoacidosis (10012632) Diabetic acidosis (10012642) Diabetic ketoacidosis (10012671) Ketoacidosis (diabetic) (10023380) Type I diabetes mellitus with ketoacidosis (10045230) Type II diabetes mellitus with ketoacidosis (10045244) |
| | Diabetic ketoacidotic<br>hyperglycaemic coma<br>(10012672) | Diabetic ketoacidotic hyperglycaemic coma (10012672)<br>Diabetic ketoacidotic hyperglycemic coma (10060579) |
| | Ketoacidosis (10023379) | Acetone breath (10000413) Breath odor ketones (10006329) Ketoacidosis (10023379) Breath odor ketones (10055425) |

<u>Note</u>: as defined in the section 11.2.4 of the protocol, diabetic ketoacidosis can be serious or non-serious AEs. Only serious ketoacidosis episodes will be considered for this analysis.

According to protocol section 11.3.3, Anticipated Adverse Device Effect (ADE) are:

- Excessive pain or discomfort from system deployment
- Excessive bleeding
- Hematoma (slight ecchymosis is a known consequence of needle skin puncture and will not be captured as an AE)
- Excessive edema from sensor and/or adhesive tape that is significant and non-resolving within 48 hours of sensor pod removal
- Excessive erythema from sensor and/or adhesive tape that is significant and non-resolving within 48 hours of sensor pod removal
- Local infection
- Sensor or introducer needle fracture during insertion/wear/removal

AEs will be coded using the MedDRA dictionary version 20.1.

# 6.4. Other endpoints and variables

# 6.4.1. Demographic data and other baseline characteristics

The following standard characteristics will be used as recorded in the eCRF:

• Baseline characteristics at V1 (i.e. age, sex, weight, height, etc.)

| Roche Diabetes Care | Statistical Analysis Plan | Page <b>22</b> / <b>64</b> |
|---------------------|---------------------------|----------------------------|
| EVERSENSE | Version 2.0 – 30/09/2020 | Page <b>22</b> / <b>64</b> |

- Diabetes history (i.e. diabetes duration, type of diabetes, usual blood glucose monitoring: capillary blood glucose or flash system, mean daily duration in hypoglycemia < 70 mg/dL, mean daily duration in hypoglycemia < 54 mg/dL, etc.)</li>
- Diabetes complications
- Last HbA1c analysis
- Diabetes Family History
- Diabetes Medication
- · Medical history diseases other than Diabetes
- Previous medications for diseases other than Diabetes
- Training at sensor insertion (D0) (arm chosen for the insertion, trained physician, etc.)
- Training to the device after randomization (at D30) for Enabled group

In addition, the following variables will be computed:

- Age (years) = (date of signed consent date of birth) / 365.25
- BMI classified according to the World Health Organization (WHO):
  - <18.5 Underweight</p>
  - 18.5 <25 Normal weight
  - 25 <30 Pre-obesity
  - o ≥30 Obesity
- Percentage of time spent in hypoglycemia < 70 mg/dL at screening and inclusion visit= (mean daily duration in hypoglycemia < 70 mg/dL (minutes) \* 100) / 1440</li>
- Percentage of time spent in hypoglycemia < 54 mg/dL at screening and inclusion visit= (mean daily duration in hypoglycemia < 54 mg/dL (minutes) \* 100) / 1440</li>
- Time since start of diabetes (years) = (date of signed consent diabetes start date) / 365.25
- Time since last blood test for HbA1c (days) = (date of screening visit date of blood test +1)
- Duration of insertion procedure (minutes) = (end time of laying strips opening time of the kit + 1)
- Duration of removal procedure (minutes) = (end time of procedure start time of procedure +1)

# 6.4.2. Follow-up data

The following data will be used as recorded in the eCRF:

- Characteristics at follow-up visit: D60, D150 and D180 (including the percentage of sensor use since the last visit, etc.)
- Training to the device at D120 for patients who switched from control to enabled group

# 6.4.3. Medical history

Medical and surgical history will be coded with the MedDRA version 20.1.

# **6.4.4.** Prior and concomitant therapies

Prior therapies are therapies which stopped before the sensor introduction. Concomitant therapies are therapies which ended on or after the sensor introduction or are ongoing at the end of the trial.

Prior and concomitant therapies will be coded with the WHO-DD version SEP 2013 format C.

#### 6.4.5. Extent of exposure

Extent of exposure will be computed as follows:

| Roche Diabetes Care | Statistical Analysis Plan | Daga 22 / 64 |
|---------------------|---------------------------|---------------------|
| EVERSENSE | Version 2.0 – 30/09/2020 | Page <b>23 / 64</b> |

- Extent of exposure (days) to investigational system = removal date of the last sensor insert date of the first sensor + 1 day.
- Extent of exposure (days), excluding period when the patient has no sensor inserted =
  [(removal date of the first sensor insert date of the first sensor) + (removal date of sensor n°X
   insert date of sensor n°X)] + 1 day

# Note:

Patient from Center died on Removal date of this sensor in place this day will be replaced with the date of the death.

Patient from Center encountered a natural ejection of the sensor. An adverse event form has been completed accordingly. Removal date of this sensor will be replaced with the resolution date of this AE.

| Roche Diabetes Care | Statistical Analysis Plan | Do 24 / 64 |
|---------------------|---------------------------|---------------------|
| EVERSENSE | Version 2.0 – 30/09/2020 | Page <b>24 / 64</b> |

# 7. DATA ANALYSIS CONSIDERATIONS

# 7.1. Statistical software

The statistical analysis will be performed using SAS° software v9.4 (or a more recent version).

# 7.2. Type I error, handling of multiplicity issues and alpha adjustment procedures

The global significance level (type I error rate) is set to  $\alpha$  = 0.05 (two-sided).

The analysis will be carried separately for each cohort. No adjustment for multiplicity is planned because analyses of both cohorts have distinct primary objective and distinct primary endpoint.

No adjustment for multiplicity with regards to multiple secondary efficacy endpoints is planned.

# 7.3. Center effect and pooling of Centers

Center effect will be included in the statistical analysis of:

- The primary endpoint of cohort 1
- The primary endpoint of cohort 2
- The secondary efficacy endpoints of cohort 1 (see section 8.6 for further details).
- The secondary efficacy endpoints of cohort 2 (see section 8.6 for further details).

For each analysis, p-value of the Center effect will be displayed. No by-center analysis is planned. Center effect will not be studied for other endpoints.

If needed (e.g. if size of some Centers is small), Centers will be pooled together according to geographic region.

Reminder: the randomization has been stratified by Center (for cohort 2) and by Center and diabetes type (for cohort 1).

# 7.4. Descriptive analyses of quantitative and qualitative variables

Continuous data will be described by the number of missing data, number of data analyzed, mean, standard deviation, median, Q1, Q3, minimum, maximum and 95% confidence interval of the mean (using the normal law).

Categorical data will be described by the number of missing data, frequencies and percentages of patients in each modality, and 95% confidence intervals (using binomial law). The percentage of patients will be calculated once missing data are excluded from the denominator.

| Roche Diabetes Care | Statistical Analysis Plan | Dogo 25 / 64 |
|---------------------|---------------------------|---------------------|
| EVERSENSE | Version 2.0 – 30/09/2020 | Page <b>25 / 64</b> |

# 7.5. Definition of baseline, time-windows and analysis periods

#### **Baseline:**

As a general rule, baseline is defined as the last available value collected prior to start of trial medication. Note that for some trial procedures this may be the value measured on the same day the trial medication was started.

# **Time-windows:**

For eCRF data, dates of visit will be used as collected in the eCRF.

For endpoints calculated with CGM data, actual dates recorded in CGM files will be used. Days will be computed using date of randomization (D30) as the reference date, for example:

- D0 = date of D30 30 days
- D30 = date of D30
- D60 = date of D30 + 30 days
- D90 = date of D30 + 60 days
- D120 = date of D30 + 90 days
- D150 = date of D30 + 120 days
- D180 = date of D30 + 150 days

Time-windows for CGM endpoints are defined as follows:

| Time-windows | Start datetime | Stop datetime[1] |
|---|---|---|
| D0-D30 | Date of visit 2 and end time of laying strips* as recorded at visit 2 (D0) + 24 hours** | Date and time of randomization recorded at D30 – 1 minute For follow-up group: date of visit D30 at 23:59. |
| D30-D60 | Date and time of randomization recorded at D30 For follow-up group: date of visit D30 at 23:59 + 1 minute. | D59 (date of visit D30 + 29 days)<br>at 23:59 |
| D60-D90 | D60 (date of visit D30 + 30 days)<br>at 00:00 | D89 (date of visit D30 + 59 days)<br>at 23:59 |
| D90-D120 | D90 (date of visit D30 + 60 days)<br>at 00:00 | D119 (date of visit D30 + 89 days) at 23:59 For control group of cohort 2: minimum date between (D119 at 23:59) and (date of switch at 23:59) |
| D120-D150 | D120 (date of visit D30 + 90 days) at 00:00 For control group of cohort 2: minimum date between (D120 at 00:00) and (date of switch at 23:59 + 1 minute) | D149 (date of visit D30 + 119 days)<br>at 23:59 |

| Roche Diabetes Care | Statistical Analysis Plan | Daga <b>36</b> / 64 |
|---------------------|---------------------------|---------------------|
| EVERSENSE | Version 2.0 – 30/09/2020 | Page <b>26 / 64</b> |

| Time-windows | Start datetime | Stop datetime[1] |
|---|---|---|
| D150-D180 | D150 (date of visit D30 + 120 days)<br>at 00:00 | Date of visit 7 and time of sensor removal*** as recorded at visit 7 (D180) |

<sup>\*</sup> If end time of laying strips is missing at visit 2, then replaced by 23:59.

[1] For each time windows, the stop datetime will be set to the date of premature discontinuation of the patient at 23:59 if it happens during this period, with date of premature discontinuation defined as the minimum between date of study withdrawal, consent withdrawal, last contact date, or death.

# 7.6. Handling of missing data and intercurrent events

# Date of birth:

| Date as collected in the CRF | Imputed date (for the analysis) |
|-------------------------------------|-------------------------------------|
| Year is complete, month is complete | Day replaced with 01. |
| Year is complete, month is missing | Day and month replaced with 01-Jul. |
| Year is missing, month is missing | Not replaced. |

# **Start date of diabetes:**

| Date as collected in the CRF | Imputed date (for the analysis) |
|---|---|
| Year is complete, month is complete, day is missing | Day replaced with 01. |
| Year is complete, month and day are missing | Day and month replaced with 01-Jul. |
| Year, month and day are missing | Not replaced. |

# **Handling of missing date for AE:**

| Onset date of AE | Imputed AE onset date (for the analysis) |
|---|---|
| Completely missing | Date of sensor insertion |
| Day is missing, month and year are filled in | If month and year are different from the first sensor insertion: |
| | Day will be replaced with first day of the month. |
| | If month and year are identical to the first sensor insertion: |
| | AE onset date will be replaced with date of first sensor insertion. |
| Day and month are | If year is different from the first sensor insertion: |
| missing, year is filled in | Day and month will be replaced with 1 <sup>st</sup> January. |

<sup>\*\*</sup> The blinded transmitter is placed 24 hours after insertion.

<sup>\*\*\*</sup> If time of sensor removal is missing at visit 7, then replaced by 00:00.

| Roche Diabetes Care | Statistical Analysis Plan | Dogo 27 / 64 |
|---------------------|---------------------------|---------------------|
| EVERSENSE | Version 2.0 – 30/09/2020 | Page <b>27 / 64</b> |

| Onset date of AE | Imputed AE onset date (for the analysis) |
|---|---|
| | If year is identical to the first sensor insertion |
| | AE onset date will be replaced with date of first sensor insertion. |

Partially or completely missing end dates of AE will not be imputed.

# Handling of missing date for sensor insertion:

| Sensor insertion date | Imputed date of sensor insertion |
|---|---|
| Completely missing | Date of first measurement for this sensor using CGM data. |
| Day is missing, month and year are filled in | If month and year are different from the first measurement for this sensor using CGM file: |
| | Day will be replaced with first day of the month. |
| | If month and year are identical to the first measurement for this sensor using CGM file: |
| | Sensor insertion date will be replaced with date of first measurement for this sensor using CGM data. |
| Day and month are missing, year is filled | If year is different from the first measurement for this sensor using CGM file: |
| in | Day and month will be replaced with 1st January. |
| | If year is identical to the first measurement for this sensor using CGM file: |
| | Sensor insertion date will be replaced with date of first measurement for this sensor using CGM data. |

# Handling of missing date for sensor removal:

| Sensor removal date | Imputed date of sensor removal |
|---|---|
| Completely missing | Date of last measurement for this sensor using CGM data. |
| Day is missing, month and year are filled in | If month and year are different from the last measurement for this sensor using CGM file: |
| | Day will be replaced with first day of the month. |
| | If month and year are identical to the last measurement for this sensor using CGM file: |
| | Sensor removal date will be replaced with date of last measurement for this sensor using CGM data. |
| Day and month are missing, year is filled | If year is different from the last measurement for this sensor using CGM file: |
| in | Day and month will be replaced with 1st January. |
| | If year is identical to the last measurement for this sensor using CGM file: |

| Roche Diabetes Care | Statistical Analysis Plan | Daga 29 / 64 |
|---------------------|---------------------------|---------------------|
| EVERSENSE | Version 2.0 – 30/09/2020 | Page <b>28 / 64</b> |

| Sensor removal date | Imputed date of sensor removal |
|---|---|
| | Sensor removal date will be replaced with date of last measurement for this sensor using CGM data. |

# Handling of intercurrent events for HbA1c (%) values:

HbA1c (%) values measured more than 30 days after the last measurement of glycemia using CGM will be excluded from the analysis (i.e. set to missing).

# Handling of missing HbA1c (%) level:

| HbA1c (%) level | Imputed value of HbA1c (%) level |
|---|---|
| D180 is missing, D120 and D0 are available | Last Observation Carried Forward (LOCF) imputation |
| D120 is missing, D180 and D0 are available | Linear interpolation |
| D120 and D180 are missing, D0 is available | Baseline Observation Carried Forward (BOCF) imputation |
| D0 is missing | No replacement, no matter if D120 and/or D180 are available |

Note: HbA1c (%) level is collected at D0, D120 and D180.

#### Handling of missing percentage of time spent in-, below- and above- target ranges:

Note: as a general rule, Method 2 + Method 3 will be used for primary analyses. Method 1 will be used for sensitivity analyses. Method 3 (only) will be used for sensitivity analyses. See Section 8.6 for further details.

# Method 1: observed cases (i.e. no replacement)

Percentages of time will be computed using all available CGM data in the specified time-window, according to the algorithm defined in section 9.2. If no CGM data is available in the specified time-window (e.g. no CGM data recorded between D90 and D120), the percentage of time spent in hypoglycemia, euglycemia and hyperglycemia will be considered as missing.

# Method 2: shift of the time-window

Assuming a specific time-window with a lower bound (L) and an upper bound (U). D is the date of measurement of the last glycemia value recorded within the time-window, and  $\Delta$  is the number of days between D and U.

- If D = U (i.e. there was no interruption of the CGM system): the percentages of time spent in-, below- and above the target range and the availability of sensor data will be computed within the (L;U) time-window.
- If D < U (i.e. there was an interruption of the CGM system): the percentages of time spent in-, below- and above the target range and the availability of sensor data will be computed within the  $(L-\Delta ; U-\Delta)$  time-window.

| Roche Diabetes Care | Statistical Analysis Plan | Daga <b>20</b> / 64 |
|---------------------|---------------------------|---------------------|
| EVERSENSE | Version 2.0 – 30/09/2020 | Page <b>29 / 64</b> |

# Note:

This method doesn't apply if no glycemia data has been recorded within the time window (L;U).

# For example:

Within the time-window D150-D180, the last available glycemia value is recorded at D170. Then, the percentages of time spent in-, below- and above the target range will be computed using all available CGM data within the D140-D170 time-window.



# Method 3: linear interpolation, LOCF and BOCF.

Percentages of time will first be computed according to the algorithm defined in section 9.2, using all available CGM data in each of the following time-windows: D0-D30, D30-D60, D60-D90, D90-D120, D120-D150 and D150-D180. If no CGM data is available in one or several time-windows, the endpoint will be imputed as follows.

1. Endpoint missing in time-window N and available in time-windows N-1 and N+1:

| D0-D30 | D30-D60 | D60-D90 | D90-D120 | D120-D150 | D150-D180 | Imputed percentage |
|---|---|---|---|---|---|---|
| Х | | Х | Х | Х | Х | Linear interpolation |
| Х | Х | | Х | Х | Х | Linear interpolation |
| Х | Х | Х | | Х | Х | Linear interpolation |
| Х | Х | Х | Х | | Х | Linear interpolation |
| Χ | · | · | Х | Х | Х | Linear interpolation |
| Χ | Х | • | • | Х | Х | Linear interpolation |
| Х | Х | Χ | | | Х | Linear interpolation |
| Х | | • | | Х | Х | Linear interpolation |
| Х | Х | • | | | Х | Linear interpolation |
| Х | • | ÷ | • | • | Х | Linear interpolation |

<sup>&</sup>quot;X": endpoint is available

# 2. Endpoint available in time-window N and missing in all subsequent N+1 time-window(s):

| D0-D30 | D30-D60 | D60-D90 | D90-D120 | D120-D150 | D150-D180 | Imputed percentage |
|---|---|---|---|---|---|---|
| Х | Х | Χ | Х | Х | • | LOCF |
| Х | Х | Х | Х | | | LOCF |
| Х | Х | Х | • | • | • | LOCF |

<sup>&</sup>quot;.": endpoint is missing (i.e. no CGM data collected during this time-window).

| Roche Diabetes Care | Statistical Analysis Plan | Dogo 20 / 64 |
|---------------------|---------------------------|---------------------|
| EVERSENSE | Version 2.0 – 30/09/2020 | Page <b>30 / 64</b> |

| D0-D30 | D30-D60 | D60-D90 | D90-D120 | D120-D150 | D150-D180 | Imputed percentage |
|---|---|---|---|---|---|---|
| Х | Х | · | · | · | · | LOCF |
| Х | | | | | | BOCF |

<sup>&</sup>quot;X": endpoint is available

<u>Note</u>: this algorithm doesn't apply to availability of CGM data (see Section 6.2.7 for computation rules of availability of CGM data).

<sup>&</sup>quot;.": endpoint is missing (i.e. no CGM data collected during this time-window).

| Roche Diabetes Care | Statistical Analysis Plan | Dogo 21 / 64 |
|---------------------|---------------------------|---------------------|
| EVERSENSE | Version 2.0 – 30/09/2020 | Page <b>31 / 64</b> |

# 8. PLANNED STATISTICAL ANALYSES

Patients will be analyzed as treated for all analyses.

# 8.1. Disposition of patients

The following will be provided by cohort, by intervention arm for the follow-up set of patients and overall:

- Number of screened patients
- Number of patients with the sensor inserted at V2 (D0)
- Number of randomized patients
- Number of patients not randomized
- Among randomized patients:
  - o Number and percentage of patients who completed the trial
  - Number and percentage of patients who prematurely discontinued from trial and reasons for withdrawal
- For cohort 2, patient randomized in control arm:
  - o Number and percentage of patients who switched to enabled arm at D120.

The following templates will be used.

| | C1 | C2 | Total |
|------------------------------------------------|-----|-----|-------|
| Patients screened | - | - | xxx |
| Patient with no sensor inserted at V2 (D0) | XXX | XXX | XXX |
| If no sensor inserted, reasons for withdrawal: | | | |
| Withdrawal of consent | XXX | XXX | XXX |
| Lost view | XXX | xxx | XXX |
| Death | XXX | XXX | XXX |
| Investigator's decision | XXX | XXX | XXX |
| Non randomization | XXX | XXX | XXX |
| Other | XXX | XXX | XXX |
| Patients with the sensor inserted at V2 (D0) | XXX | XXX | XXX |
| If sensor inserted, patients not randomized | XXX | xxx | XXX |
| Withdrawal of consent | XXX | XXX | XXX |
| Lost view | XXX | XXX | XXX |
| Death | XXX | XXX | XXX |
| Investigator's decision | XXX | xxx | XXX |
| Non randomization | XXX | XXX | XXX |
| Other | XXX | xxx | XXX |

| Roche Diabetes Care | Statistical Analysis Plan | Page 22 / 64 |
|---------------------|---------------------------|---------------------|
| EVERSENSE | Version 2.0 – 30/09/2020 | Page <b>32 / 64</b> |

| | Cohort 1 | | |
|---------------------------|-------------|-------------|------------|
| | Enabled Arm | Control arm | Total |
| Patients randomized | XXX | XXX | XXX |
| Among randomized patients | | | |
| trial completed | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| prematurely discontinued | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Reasons for withdrawal: | | | |
| Withdrawal of consent | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Lost view | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Death | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Investigator's decision | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Non randomization | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Other | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

| | Cohort 2 | | |
|---|---|---|---|
| | Enabled Arm | Control arm | Total |
| Patients randomized | XXX | xxx | xxx |
| Patients not randomized | XXX | xxx | xxx |
| Included in the follow-up set | XXX | xxx | XXX |
| Not included in the follow-up set | XXX | XXX | XXX |
| Among randomized patients | | | |
| trial completed | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| prematurely discontinued | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Patients who switched to enabled arm at D120 | - | xx (xx.x%) | xx (xx.x%) |
| Reasons for withdrawal: | | | |
| Withdrawal of consent | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Lost view | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Death | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Investigator's decision | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Non randomization | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Other | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

# In addition, the following data will be provided:

- Date of first patient screened (i.e. date of signed consent)
- Date of first patient with inserted sensor
- Date of last patient with inserted sensor

| Roche Diabetes Care | Statistical Analysis Plan | Page 22 / 64 |
|---------------------|---------------------------|---------------------|
| EVERSENSE | Version 2.0 – 30/09/2020 | Page <b>33 / 64</b> |

- Date of first patient randomized
- Date of last patient randomized
- Date of last patient out (i.e. last visit performed)
- Overall study duration (days) = date of last patient last visit date of first patient screened +1

#### 8.2. Protocol deviations

Major protocol deviations will be described on all randomized patients, by intervention arm and overall

Pre-specified major protocol deviations categories are:

- Inclusion criteria not met and/or exclusion criteria met [1]
- Informed consent not available or given too late
- Patient selected in the wrong cohort (e.g. Cohort 1 instead of Cohort 2)
- Patient randomized in the wrong intervention arm (e.g. Enabled instead of Control)
- Use of prohibited (prior and / or concomitant) medication
- Missing primary endpoint (i.e. missing CGM data or insufficient availability of CGM data)

Further categories of major protocol deviations can be defined during the data review meeting. List of major protocol deviations will be finalized in the data review minutes and approved by the Sponsor.

[1] Note: Exclusion criterion 3 is not collected for patients selected before March 29th, 2019. Definition of exclusion criterion 5 and criterion 7 is not the same for patients selected before and after March 29<sup>th</sup>, 2019.

# 8.3. Analysis sets and cohorts analyzed

Frequency and percentage of patients included in each analysis sets defined in Section 5 will be provided by treatment group and overall by cohort, by intervention arm and overall.

# 8.4. Demographic data and baseline characteristics, including medical history and therapies

# 8.4.1. Analysis of demographic data and other baseline characteristics

Descriptive analyses will be provided by cohort and overall on the Safety Set.

In addition, percentage of time spent in hypoglycemia <54 mg/dL as collected in the eCRF at visit V1 (i.e. screening) for Cohort 1 and at visit V3 (i.e. D30) for Cohort 2 according to the usual glucose monitoring system will be compared to percentage of time spent in hypoglycemia <54 mg/dL as computed with CGM data between D0-D30 using a (non parametric) Wilcoxon test. This analysis will be provided by cohort, on the safety set. The following templates will be used.

| Roche Diabetes Care | Statistical Analysis Plan | Daga 24 / 64 |
|---------------------|---------------------------|---------------------|
| EVERSENSE | Version 2.0 – 30/09/2020 | Page <b>34 / 64</b> |

| | | Cohort 1 | |
|---|---|---|---|
| | Statistical<br>test | Data collected in eCRF at visit 1 (D0) [1] (N=xxx) | Data computed with CGM data between D0-D30 [2] (N=x) |
| Percentage of time<br>spent in hypoglycemia<br><54mg/dL:<br>N<br>Mean (SD)<br>Median<br>Q1; Q3<br>Min; Max | Wilcoxon<br>p = x.xxx | xxx<br>xx.x (xx.x)<br>xx.x<br>xx.x; xx.x<br>xx.x; xx.x | xxx<br>xx.x (xx.x)<br>xx.x<br>xx.x; xx.x<br>xx.x; xx.x |

<sup>[1]</sup> computed as (100 \* daily mean time (minutes) spent below 54 mg/dL during the last 28 days according to usual glucose monitoring system and reported in the eCRF by investigators) / 1440.

<sup>[2]</sup> computed using CGM data from Eversense system, according to algorithm defined in SAP.

| | | Cohort 2 | |
|---|---|---|---|
| | Statistical<br>test | Data collected in eCRF at visit 3 (D30) [1] (N=xxx) | Data computed with CGM data between D0-D30 [2] (N=x) |
| Percentage of time<br>spent in hypoglycemia<br><54mg/dL:<br>N<br>Mean (SD)<br>Median<br>Q1; Q3<br>Min; Max | Wilcoxon p = x.xxx | xxx<br>xx.x (xx.x)<br>xx.x<br>xx.x; xx.x<br>xx.x; xx.x | xxx<br>xx.x (xx.x)<br>xx.x<br>xx.x; xx.x<br>xx.x; xx.x |

<sup>[1]</sup> computed as  $(100 * daily mean time (minutes) spent below 54 mg/dL between visit V2 (i.e. D0, _insertion) and visit V3 (i.e. D30, randomization) according to usual glucose monitoring system and reported in the eCRF by investigators) / 1440. [2] computed using CGM data from Eversense system, according to algorithm defined in SAP.$ 

# 8.4.2. Analysis of follow-up data

Descriptive analyses will be provided by cohort and overall on the Safety Set.

# 8.4.3. Analysis of Medical and surgical history

Descriptive analyses will be provided by cohort and overall on the Safety Set.

Medical and surgical history will be analyzed by MedDRA System Organ Class (SOC) and Preferred Term (PT). The SOC will be sorted by descending frequency and PT will be sorted by descending frequency (within SOC, on «total» column).

# 8.4.4. Analysis of Prior and concomitant therapies

Descriptive analyses will be provided by cohort and overall on the Safety Set.

Prior and concomitant therapies will be analyzed separately, by WHO-DD preferred name and ATC3. The ATC3 will be sorted by descending frequency and WHO-DD preferred names will be sorted by descending frequency (within ATC3, on « total » column).

| Roche Diabetes Care | Statistical Analysis Plan | Daga 25 / 64 |
|---------------------|---------------------------|---------------------|
| EVERSENSE | Version 2.0 – 30/09/2020 | Page <b>35 / 64</b> |

# 8.5. Analysis of extent of exposure and treatment compliance

The criteria defined in section 6.4.5 will be described by cohort, intervention arm and overall on the Safety Set.

# 8.6. Efficacy analysis

As a general rule, statistical models for cohort 1 will include center and diabetes type as stratification variables and HbA1c (%) at D0 as baseline covariate. Statistical models for cohort 2 will include center as stratification variable and HbA1c (%) as baseline covariate.

# 8.6.1. Analysis of the primary efficacy endpoint

# 8.6.1.1. Cohort 1: HbA1c (%) at D180

#### **Descriptive analysis:**

A descriptive analysis of HbA1c (%) at D180 will be provided by intervention arm on the FAS (with handling of intercurrent events and missing HbA1c values). The following template will be used.

| | Cohort 1 | |
|---------------------------|--------------|-------------------|
| | Enabled arm | Control arm |
| | N=XXX | N=XXX |
| HbA1C (%) at baseline | | |
| (screening visit) | | |
| Non-missing | XX | XX |
| Missing | XX | xx |
| Mean (±SD) | xx.x (±xx.x) | $xx.x (\pm xx.x)$ |
| 95% CI | [xx.x;xx.x] | [xx.x;xx.x] |
| Median | XX.X | XX.X |
| Q1-Q3 | [xx.x;xx.x] | [xx.x;xx.x] |
| Min-Max | [xx.x;xx.x] | [xx.x;xx.x] |
| HbA1C (%) at D180 | | |
| Non-missing | XX | xx |
| Missing | XX | XX |
| Mean (±SD) | xx.x (±xx.x) | $xx.x (\pm xx.x)$ |
| 95% CI | [xx.x;xx.x] | [xx.x;xx.x] |
| Median | XX.X | XX.X |
| Q1-Q3 | [xx.x;xx.x] | [xx.x;xx.x] |
| Min-Max | [xx.x;xx.x] | [xx.x;xx.x] |
| Change in HbA1C (%) | | |
| between baseline and D180 | | |
| Non-missing | XX | xx |
| Missing | XX | xx |
| Mean (±SD) | xx.x (±xx.x) | $xx.x (\pm xx.x)$ |
| 95% CI | [xx.x;xx.x] | [xx.x;xx.x] |
| Median | XX.X | XX.X |
| Q1-Q3 | [xx.x;xx.x] | [xx.x;xx.x] |
| Min-Max | [xx.x;xx.x] | [xx.x;xx.x] |

#### Main analysis (parametric model):

The analysis of the primary endpoint for cohort 1 will be an analysis of covariance (ANCOVA) comparing the HbA1c (%) at D180 visit between treatment arms. The statistical model will include randomization arm, center and diabetes type as fixed classification effects and HbA1c (%) at D0 as baseline covariates. Adjusted means with their 95% CI will be provided. P-values of each effects and covariates will be displayed. Intercurrent events and missing HbA1c values will be handled as described in Section 7.6. The primary analysis will be provided on the FAS. The following template will be used.
| Roche Diabetes Care | Statistical Analysis Plan | Daga 36 / 64 |
|---------------------|---------------------------|---------------------|
| EVERSENSE | Version 2.0 – 30/09/2020 | Page <b>36 / 64</b> |

| Enabled arm Control arm Difference N=XXX N=XXX (Enabled - control) HbAlC (%) at D180 | | Cohort 1 | | |
|---|---|---|---|---|
| HbA1C (%) at D180 xx.x xx.x xx.x Adjusted mean xx.x xx.x xx.x 95% CI [xx.x;xx.x] [xx.x;xx.x] [xx.x;xx.x] | | Enabled arm | Control arm | Difference |
| Adjusted mean xx.x xx.x xx.x 95% CI [xx.x;xx.x] [xx.x;xx.x] [xx.x;xx.x] | | N=XXX | N=XXX | (Enabled - control) |
| | Adjusted mean<br>95% CI | | - | [xx.x;xx.x] |

From an ANCOVA model including Center (p=0.xxx) and diabetes type (p=0.xxx) as fixed classification effect, HbA1c (%) level at baseline (p=0.xxx) as baseline covariates.

Note: the primary endpoint for Cohort 1 is HbAlC (%) at D180. Note: HbAlC (%) at D180 is a secondary endpoint for Cohort 2.

The same analysis will be provided for the absolute change in HbA1c (%) from baseline to D180. The following template will be used.

| | Cohort 1 | | |
|---|---|---|---|
| | Enabled arm | Control arm | Difference |
| | N=XXX | N=XXX | (Enabled - control) |
| Change in HbA1C (%) | | | |
| between baseline | | | |
| and D180 | | | |
| Adjusted mean | xx.x | XX.X | XX.X |
| 95% CI | [xx.x;xx.x] | [xx.x;xx.x] | [xx.x;xx.x] |
| p value | | | p=0.xx |
| From an ANCOVA model | including Center | (p=0.xxx) and $(p=0.xxx)$ | diabetes type $(p=0.xxx)$ |

From an ANCOVA model including Center (p=0.xxx) and diabetes type (p=0.xxx) as fixed classification effect, HbAlc (%) level at baseline (p=0.xxx) as baseline covariates.

Note: normality of distribution will be studied using a histogram with the normal probability density curve. Distribution of HbA1c (%) at D180 in Cohort 1 may be skewed, due to inclusion criterion #3 (i.e. HbA1c level at baseline > 8%). The gamma distribution will be studied using a histogram with the gamma probability density curve. If applicable, the ANCOVA models described above will be replaced by a Generalized Linear Models (GLM) using a Gamma distribution and a LOG link function. The statistical model will include randomization arm, center and diabetes type as fixed classification effects and HbA1c (%) at D0 as baseline covariates. Adjusted means with their 95% CI will be provided. P-values of each effects and covariates will be displayed. The same templates will be used.

### Sensitivity analysis #1: (non-parametric model)

The primary endpoint will be classified as follows: less than 6%, 6-<7%, 7-<8%, 8-<9% 9-<10%, 10% and more. A Generalized Linear Model (GLM) for ordinal data with multinomial distribution and a cumulative link will be used. The cumulative logit model will include randomization arm, center, diabetes type and HbA1c (%) at D0 as baseline covariates. Log odds ratio will be exponentiated to form odds ratio estimates. This model will be used to compute odds ratio with their 95% CI and corresponding p-value. The primary analysis will be provided on the FAS with method 3 ("linear interpolation, LOCF and BOCF", cf. Section 7.6) for handling of missing data.

The following template will be used.

| Roche Diabetes Care | Statistical Analysis Plan | Daga 27 / 64 |
|---------------------|---------------------------|---------------------|
| EVERSENSE | Version 2.0 – 30/09/2020 | Page <b>37 / 64</b> |

| | Coho | ort 2 |
|---|---|---|
| | Enabled | Control |
| | N=XXX | N=XXX |
| HbA1C (%) at D180 - N(%) | | |
| Less than 6% | xx ( xx.x) | xx ( xx.x) |
| 6-7% | xx ( xx.x) | xx ( xx.x) |
| 7-8% | xx ( xx.x) | xx ( xx.x) |
| 8-9% | xx ( xx.x) | xx ( xx.x) |
| 9-10% | xx ( xx.x) | xx ( xx.x) |
| More than 10% | xx ( xx.x) | xx ( xx.x) |
| Adjusted odds ratio (Enabled vs Control) [1] | xx.x | _ |
| 95% CI | [xx.x;xx.x] | |
| p-value | p=0.xxx | |
| [1] From a cumulative logit model including center (p=0.xxx) as fixed | | |
| classification effect and HbA1c (%) level at baseline (p=0.xxx) as covariate. | | |

<u>Note</u>: an odds ratio "x" statistically greater than 1.0 (i.e. 95% low confidence limit > 1.0) will indicate odds of Enabled group being in lower HbA1c categories is "x" times the odds of Control group being in lower HbA1c categories. Since the lower categories represent the more favorable results, this would indicate that Enabled group is significantly better than Control group.

### Sensitivity analysis #2:

The main analysis and descriptive analysis described above will be provided on the FAS on all observed cases (i.e. without handling of intercurrent events and without replacement of missing data).

### Sensitivity analysis #3:

The main analysis and descriptive analysis described above will be provided on the Per Protocol Set. Intercurrent events and missing HbA1c values will be handled as described in Section 7.6.

| Roche Diabetes Care | Statistical Analysis Plan | Dogo 39 / 64 |
|---------------------|---------------------------|---------------------|
| EVERSENSE | Version 2.0 – 30/09/2020 | Page <b>38 / 64</b> |

## 8.6.1.2. Cohort 2: Percentage of time in hypoglycemia <54mg/dL between D90 visit and D120 visit

### **Descriptive analysis:**

A descriptive analysis, both continuous and qualitative (i.e. by classes of 1%), of the percentage of time spent in hypoglycemia <54mg/dL between D90 and D120 and at baseline (i.e. between D0 and D30) will be provided by cohort and by intervention arm, on the FAS with method 3 ("linear interpolation, LOCF and BOCF", cf. Section 7.6) for handling of missing data..

The following template will be used.

| | Cohort 2 | |
|---|---|---|
| | Enabled | Control |
| | N=XXX | N=XXX |
| Percentage of time spent in hypoglycemia | 17 712121 | 17 212121 |
| <pre>&lt;54mg/dL between D0 and D30</pre> | | |
| Non-missing | xx | XX |
| Missing | XX | XX |
| Mean (±SD) | xx.x (±xx.x) | xx.x (±xx.x) |
| 95% CI | [xx.x;xx.x] | [xx.x;xx.x] |
| Median | XX.X | XX.X |
| 01-03 | [xx.x;xx.x] | [xx.x;xx.x] |
| Min-Max | [xx.x;xx.x] | [xx.x;xx.x] |
| Less than 1% | xx (xx.x) | xx (xx.x) |
| 1-<2% | xx (xx.x) | xx (xx.x) |
| 2-<3% | xx (xx.x) | xx (xx.x) |
| 3-<4% | xx (xx.x) | xx (xx.x)<br>xx (xx.x) |
| 4-<5% | xx (xx.x)<br>xx (xx.x) | xx (xx.x)<br>xx (xx.x) |
| 5-<6% | xx (xx.x) | xx (xx.x) |
| 6-<7% | xx (xx.x) | xx (xx.x) |
| 7-<8% | xx (xx.x) | xx (xx.x) |
| 8-<9% | xx (xx.x) | xx (xx.x) |
| 9-<10% | xx (xx.x) | xx (xx.x) |
| 10-<11% | xx (xx.x) | xx (xx.x) |
| Etc.% | | |
| Percentage of time spent in hypoglycemia | | |
| <54mg/dL between D90 and D120 | | |
| Non-missing | XX | XX |
| Missing | XX | XX |
| Mean (±SD) | xx.x (±xx.x) | xx.x (±xx.x) |
| 95% CI | [xx.x;xx.x] | [xx.x;xx.x] |
| Median | XX.X | XX.X |
| Q1-Q3 | [xx.x;xx.x] | [xx.x;xx.x] |
| Min-Max | [xx.x;xx.x] | [xx.x;xx.x] |
| Less than 1% | xx (xx.x) | xx (xx.x) |
| 1-<2% | xx (xx.x) | xx (xx.x) |
| 2-<3% | xx (xx.x) | xx (xx.x) |
| 3-<4% | xx (xx.x) | xx (xx.x) |
| 4-<5% | xx (xx.x) | xx (xx.x) |
| 5-<6% | xx (xx.x) | xx (xx.x) |
| 6-<7% | xx (xx.x) | xx (xx.x) |
| 7-<8% | xx (xx.x) | xx (xx.x) |
| 8-<9% | xx (xx.x) | xx (xx.x) |
| 9-<10% | xx (xx.x) | xx (xx.x) |
| 10-<11% | xx (xx.x) | xx (xx.x) |
| Etc.% | | |

Note: the primary endpoint for Cohort 2 is the percentage of time in hypoglycemia. Note: Percentage of time in hypoglycemia is a secondary endpoint for Cohort 1. Note: Percentage of time in hypoglycemia between D0 and D30 is the baseline value.

| Roche Diabetes Care | Statistical Analysis Plan | Dogo 20 / 64 |
|---------------------|---------------------------|---------------------|
| EVERSENSE | Version 2.0 – 30/09/2020 | Page <b>39 / 64</b> |

### Main analysis (parametric model):

The analysis of the primary endpoint for cohort 2 will be an analysis of covariance (ANCOVA) comparing the percentage of time spent in hypoglycemia <54mg/dL between D90 visit and D120 visit between treatment arms. The statistical model will include randomization arm and center as fixed classification effects and the level of hypoglycemia at baseline (i.e. percentage of time spent in hypoglycemia <54 mg/dl between D0 visit and D30 visit) as baseline covariates. Adjusted means with their 95% CI will be provided. P-values of each effects and covariates will be displayed. Missing values will be handled as described in Section 7.6 using method 3 "linear interpolation, LOCF and BOCF". The primary analysis will be provided on the FAS.

The following template will be used.

| | | Cohort | . 2 |
|---|---|---|---|
| | Enabled | Control | Difference |
| | N=XXX | N=XXX | (Enabled - control) |
| Percentage of time in hypoglycemia <54mg/dL between D90 and D120 | | | |
| Adjusted mean | XX.X | XX.X | XX.X |
| 95% CI | [xx.x;xx.x] | [xx.x;xx.x] | [xx.x;xx.x] |
| p value | | | p=0.xxx |
| From an ANCOVA model including Center | (p=0.xxx) as | fixed class: | ification effect, time |
| spent in hypoglycemia <54 mg/dl from | n DO visit to | D30 visit | (p=0.xxx) as baseline |
| covariate. | | | |

<u>Note</u>: Normality of distribution will be studied using a histogram with the normal probability density curve.

### Sensitivity analysis #1 (non-parametric model):

The primary endpoint will be classified as follows: less than 1%, 1-<2%, 2-<3%, etc., 9-<10%, 10% and more. A Generalized Linear Model (GLM) for ordinal data with multinomial distribution and a cumulative link will be used. The cumulative logit model will include randomization arm, center and percentage of time spent <54mg/dL from D0 to D30 as covariates. Log odds ratio will be exponentiated to form odds ratio estimates. This model will be used to compute odds ratio with their 95% CI and corresponding p-value. The primary analysis will be provided on the FAS with method 3 ("linear interpolation, LOCF and BOCF", cf. Section 7.6) for handling of missing data.

The following template will be used.

| | Coho | rt 2 |
|---|---|---|
| | Enabled | Control |
| | N=XXX | N=XXX |
| Percentage of time in hypoglycemia <54mg/dL | | |
| between D90 and D120 - N(%) | | |
| Less than 1% | xx ( xx.x) | xx ( xx.x) |
| 1-2% | xx ( xx.x) | xx ( xx.x) |
| 2-3% | xx ( xx.x) | xx ( xx.x) |
| 3-4% | xx ( xx.x) | xx ( xx.x) |
| 4-5% | xx ( xx.x) | xx ( xx.x) |
| 5-6% | xx ( xx.x) | xx ( xx.x) |
| 6-7% | xx ( xx.x) | xx ( xx.x) |
| 7-8% | xx ( xx.x) | xx ( xx.x) |
| 8-9% | xx ( xx.x) | xx ( xx.x) |
| 9-10% | xx ( xx.x) | xx ( xx.x) |
| More than 10% | xx ( xx.x) | xx ( xx.x) |
| Adjusted odds ratio (Enabled vs Control) [1] | XX.X | = |
| 95% CI | [xx.x;xx.x] | |
| p-value | p=0.xxx | |
| [1] From a cumulative logit model including center | r (p=0.xxx) as f | ixed |
| classification effect and percentage of time spen- | t <54mg/dL from | D0 to D30 |
| (p=0.xxx) as baseline covariate. | | |

<u>Note</u>: an odds ratio "x" statistically greater than 1.0 (i.e. 95% low confidence limit > 1.0) will indicate odds of Enabled group being in lower percentage of time categories is "x" times the odds of Control group being in lower percentage of time categories. Since the lower categories represent the more favorable percentage of time results, this would indicate that Enabled group is significantly better than Control group.

### **Sensitivity analysis #2:**

The main analysis and descriptive analysis will be provided on the FAS using method 1 (observed cases, no replacement) for handling of missing data.

### **Sensitivity analysis #3:**

The main analysis and descriptive analysis will be provided on the FAS, using method 2 (shift of the time-window) and method 3 (linear interpolation, LOCF and BOCF) for handling of missing data.

#### **Sensitivity analysis #4:**

A (non-parametric) rank-ANCOVA will be performed on the FAS with method 3 (linear interpolation, LOCF and BOCF) for handling of missing data. Rank transformation will be applied to the primary endpoint. The same ANCOVA model described above will be run on the rank-transformed primary endpoint. Only p-values will be displayed, as the computed mean values and confidence intervals are not interpretable. The purpose of this sensitivity analysis is to check robustness of the primary analysis, if normality of distribution of the primary endpoint is rejected.

The following template will be used.

| Rank-ANCOVA model for percentage of time spent in hypoglycemia | <54mg/dL |
|---|---|
| between D90 and D120 | |
| Treatment arm effect: | p=0.xxx |
| Center effect: | p=0.xxx<br>p=0.xxx |
| Time in hypoglycemia <54 mg/dl from DO visit to D30 visit effect | p=0.xxx |

| Roche Diabetes Care | Statistical Analysis Plan | Page 41 / 64 |
|---------------------|---------------------------|---------------------|
| EVERSENSE | Version 2.0 – 30/09/2020 | Page <b>41 / 64</b> |

### **Sensitivity analysis #5:**

A (non-parametric) Wilcoxon-Mann-Whitney test will be performed on the FAS with method 3 (linear interpolation, LOCF and BOCF) for handling of missing data.

The following template will be used:

| | | Cohort 2 | |
|---|---|---|---|
| | | Enabled | Control |
| | | N=XXX | N=XXX |
| Percentage of time spent in hypoglycemia | | | |
| <54mg/dL between D90 and D120 | | | |
| Non-missing | | XX | XX |
| Missing | | XX | XX |
| Median | Wilcoxon | XX.X | XX.X |
| Q1-Q3 | p=0.xxx | [xx.x;xx.x] | [xx.x;xx.x] |
| Min-Max | | [xx.x;xx.x] | [xx.x;xx.x] |

### Sensitivity analysis #6:

The main analysis and descriptive analysis described above will be provided on the Per Protocol Set. Missing values will be handled as described in Section 7.6 using method 3 "linear interpolation, LOCF and BOCF".

### 8.6.2. Analysis of the secondary efficacy endpoints

### 8.6.2.1. Safety of the insertion and removal procedures and safety of the device

A descriptive analysis of pre-specified AEs listed in section 6.2.1 will be provided by cohort and by intervention arm, on the FAS.

The following template will be used.

| | Cohort 1 | | |
|---|---|---|---|
| Pre-specified AEs which occurred after sensor insertion | Control<br>N=xxx | Enabled<br>N=xxx | Total<br>N=xxx |
| Infection, local or systemic | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) |
| Excessive bleeding | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) |
| Edema or swelling | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) |
| Scar formation and/or Keloid | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) |
| Skin irritation and/or redness | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) |
| Nerve damage causing tingling, numbness, pain or weakness | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) |
| Puritis (itching of the incision while healing) | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) |
| Discoloration of skin | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) |
| Hematoma formation | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) |
| Burning sensation and/or pain | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) |
| Device migration | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) |

The same template will be used for:

• Cohort 1: pre-specified AEs which occurred after sensor removal

| Roche Diabetes Care | Statistical Analysis Plan | Dogo 42 / 64 |
|---------------------|---------------------------|---------------------|
| EVERSENSE | Version 2.0 – 30/09/2020 | Page <b>42 / 64</b> |

- Cohort 1: pre-specified AEs which didn't occur after sensor insertion or removal
- Cohort 2: pre-specified AEs which occurred after sensor insertion
- Cohort 2: pre-specified AEs which occurred after sensor removal
- Cohort 2: pre-specified AEs which didn't occur after sensor insertion or removal

### 8.6.2.2. Analysis of percentage of time spent in the [70mg/dL-180mg/dL] glucose range

Time in range [70mg/dL-180mg/dL] of glucose values from D150 to D180.

This endpoint will be analyzed as described for the primary analysis of the cohort 2 primary endpoint, i.e. descriptive analysis and ANCOVA model on the FAS with method 3 (linear interpolation, LOCF and BOCF) for handling of missing data.

The same analysis will be provided for cohort 1.

Time in range [70mg/dL-180mg/dL] of glucose values from D90 to D120.

This endpoint will be analyzed as described for the primary analysis of the cohort 2 primary endpoint, i.e. descriptive analysis and ANCOVA model on the FAS with method 3 (linear interpolation, LOCF and BOCF) for handling of missing data.

The same analysis will be provided for cohort 1.

### 8.6.2.3. Analysis of percentage of time spent in hypoglycemia and hyperglycemia

- Time in hypoglycemia (<70mg/dL) from D150 to D180</li>
- Time in hypoglycemia (<70mg/dL) from D90 to D120</li>
- Time in hypoglycemia (<54mg/dL) from D150 to D180</li>
- Time in hypoglycemia (<54mg/dL) from D90 to D120</li>
- Time in hyperglycemia (>180mg/dL) from D150 to D180
- Time in hyperglycemia (>180mg/dL) from D90 to D120
- Time in hyperglycemia (>250mg/dL) from D150 to D180
- Time in hyperglycemia (>250mg/dL) from D90 to D120

These endpoints will be analyzed as described for the primary analysis of the cohort 2 primary endpoint, i.e. descriptive analysis and ANCOVA model on the FAS with method 3 (linear interpolation, LOCF and BOCF) for handling of missing data.

The same analysis will be provided for cohort 1.

## 8.6.2.4. Analysis of glucose variability estimated with coefficient of variation calculated by 24h as ratio of standard deviation to mean daily glucose

#### 8.6.2.4.1. Analysis of Coefficient of Variation

CV (%) measured from D90 to D120 and CV measured from D150 to D180 will be analyzed as described for the primary analysis of the cohort 2 primary endpoint, i.e. descriptive analysis and ANCOVA model on the FAS with method 3 (linear interpolation, LOCF and BOCF) for handling of missing data.

| Roche Diabetes Care | Statistical Analysis Plan | Page 42 / 64 |
|---------------------|---------------------------|---------------------|
| EVERSENSE | Version 2.0 – 30/09/2020 | Page <b>43 / 64</b> |

The following template will be used for the ANCOVA.

| | Cohort 2 | | |
|---|---|---|---|
| | Enabled | Control | Difference |
| | N=XXX | N=XXX | (Enabled - control) |
| CV (%) between D90 and D120<br>Adjusted mean | | | |
| 95% CI | XX.X | XX.X | XX.X |
| p value | [xx.x;xx.x] | [xx.x;xx.x] | [xx.x;xx.x] |
| | | | p=0.xxx |
| From an ANCOVA model including Center (%) from D0 to D30 visit (p=0.xxx) as | - | | ication effect and CV |

The same analysis will be provided for cohort 1.

### Analysis of binary CV endpoints (<36, ≥36%):

Binary endpoints (i.e. CV measured from D90 to D120 < 36% and CV measured from D150 to D180 < 36%) will be compared between treatment groups using a logistic regression model including randomization arm, center, diabetes type and HbA1c (%) at D0 as baseline covariates. This model will be used to compute odds ratio with their 95% CI and corresponding p-value. The analysis will be provided on the FAS with method 3 ("linear interpolation, LOCF and BOCF", cf. Section 7.6) for handling of missing data.

The following template will be used.

| | Cohort 1 | |
|---|---|---|
| | Enabled | Control |
| | N=XXX | N=XXX |
| CV (%) from D90 to D120- N(%) | | |
| < 36% | xx ( xx.x) | xx ( xx.x) |
| >=36% | xx ( xx.x) | xx ( xx.x) |
| Adjusted odds ratio (Enabled vs Control) [1] | XX.X | - |
| 95% CI | [xx.x;xx.x] | |
| p-value | p=0.xxx | |
| [1] From a logistic model including center (p=0.xxx) and diabetes type | | |
| (p=0.xxx) as fixed classification effects and HbA1c (%) level at baseline | | |
| (p=0.xxx) as covariate. | | |

### 8.6.2.4.2. Analysis of Blood Glucose Indexes

LBGI, HBGI and BGRI measured from D90 to D120 and measured from D150 to D180 will be analyzed as described above for the analysis of Coefficient of Variation (see section above).

### 8.6.2.5. Analysis of sensor life

A descriptive analysis will be provided by cohort and by intervention arm, on the FAS.

The following templates will be used.

| Roche Diabetes Care | Statistical Analysis Plan | Dago 44 / 64 |
|---------------------|---------------------------|---------------------|
| EVERSENSE | Version 2.0 – 30/09/2020 | Page <b>44 / 64</b> |

| | Cohort 1 | | |
|---|---|---|---|
| | Control | Enabled | Total |
| | N=XXX | N=XXX | N=XXX |
| Lifespan (days) for the first sensor: | | | |
| Non-missing | XX | XX | XX |
| Missing | XX | XX | XX |
| Mean (±SD) | $xx.x (\pm xx.x)$ | $xx.x (\pm xx.x)$ | xx.x (±xx.x) |
| 95% CI | [xx.x;xx.x] | [xx.x;xx.x] | [xx.x;xx.x] |
| Median | XX.X | XX.X | XX.X |
| Q1-Q3 | [xx.x;xx.x] | [xx.x;xx.x] | [xx.x;xx.x] |
| Min-Max | [xx.x;xx.x] | [xx.x;xx.x] | [xx.x;xx.x] |
| Patients having first sensor operating | | | |
| at D150 | | | |
| Yes [n (%)] | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No [n (%)] | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Patients having first sensor operating | | | |
| at D180 | | | |
| Yes [n (%)] | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| No [n (용)] | xx (xx.x) | xx (xx.x) | xx (xx.x) |

| | Cohort 1 | | |
|---|---|---|---|
| | Control | Enabled | Total |
| 27 1 6 | N=XXX | N=XXX | N=XXX |
| Number of sensors used between DO | | | |
| and D180 | XX | XX | XX |
| Non-missing | XX | XX | XX |
| Missing | xx.x (±xx.x) | $xx.x (\pm xx.x)$ | xx.x (±xx.x) |
| Mean (±SD) | [xx.x;xx.x] | [xx.x;xx.x] | [xx.x;xx.x] |
| 95% CI | XX.X | XX.X | XX.X |
| Median | [xx.x;xx.x] | [xx.x;xx.x] | [xx.x;xx.x] |
| Q1-Q3 | [xx.x;xx.x] | [xx.x;xx.x] | [xx.x;xx.x] |
| Min-Max | | | |
| Number of sensors used Between DO and D180 - N(%) [95%CI] 1 sensor | xx (xx.x)<br>[xx.x;xx.x] | xx (xx.x)<br>[xx.x;xx.x] | xx (xx.x)<br>[xx.x;xx.x] |
| 2 sensors | xx (xx.x)<br>[xx.x;xx.x] | xx (xx.x)<br>[xx.x;xx.x] | xx (xx.x)<br>[xx.x;xx.x] |
| 3 sensors | xx (xx.x)<br>[xx.x;xx.x] | xx (xx.x)<br>[xx.x;xx.x] | xx (xx.x)<br>[xx.x;xx.x] |
| 4 sensor<br>s () | xx (xx.x)<br>[xx.x;xx.x] | xx (xx.x)<br>[xx.x;xx.x] | xx (xx.x)<br>[xx.x;xx.x] |

Same template for number of sensors used between D0-D120, and between D30-D180.

| Roche Diabetes Care | Statistical Analysis Plan | Do 45 / 64 |
|---------------------|---------------------------|---------------------|
| EVERSENSE | Version 2.0 – 30/09/2020 | Page <b>45 / 64</b> |

A Kaplan-Meier plot of the lifespan for the first sensor will be provided (overall) on the FAS. The 95% confidence limits of the survival curve will be displayed. Confidence interval will be computed using LOG-LOG transformation.

Reminder of endpoint's definition (see section 6.2.5):

Lifespan (days) for the first sensor = Date of the last glucose measurement by the sensor –
date of the first glucose measurement by the sensor + 1

### Censoring:

- Patients with first sensor removed at D180 visit will be censored to the date of D180 visit.
- Patients with missing data (i.e. no CGM records) are excluded from the FAS.
- No other censoring rules is defined.

The following template will be used.



### 8.6.2.6. Analysis of transmitter wear time

A descriptive analysis will be provided by cohort and by intervention arm, on the FAS. This endpoint will be analyzed using the same template as for the previous criterion.

| Roche Diabetes Care | Statistical Analysis Plan | Dogo 46 / 64 |
|---------------------|---------------------------|---------------------|
| EVERSENSE | Version 2.0 – 30/09/2020 | Page <b>46 / 64</b> |

## 8.6.2.7. Analysis of availability of sensor data

A descriptive analysis will be provided by cohort and by intervention arm, on the FAS.

The following template will be used.

| | | Cohort 1 | |
|---|---|---|---|
| | Control | Enabled | Total |
| | N=XXX | N=XXX | N=XXX |
| Availability of sensor data between D0 | | | |
| and D30: | | | |
| Non-missing | XX | XX | XX |
| Missing | XX | XX | XX |
| Mean (±SD) | $xx.x (\pm xx.x)$ | xx.x (±xx.x) | xx.x (±xx.x) |
| 95% CI | [xx.x;xx.x] | [xx.x;xx.x] | [xx.x;xx.x] |
| Median | XX.X | XX.X | XX.X |
| Q1-Q3 | [xx.x;xx.x] | [xx.x;xx.x] | [xx.x;xx.x] |
| Min-Max | [xx.x;xx.x] | [xx.x;xx.x] | [xx.x;xx.x] |
| [] | [] | [] | [] |
| Availability of sensor data between DO | | | |
| and D180 (or last visit): | | | |
| Non-missing | XX | XX | XX |
| Missing | XX | XX | XX |
| Mean (±SD) | $xx.x (\pm xx.x)$ | $xx.x (\pm xx.x)$ | $xx.x (\pm xx.x)$ |
| 95% CI | [xx.x;xx.x] | [xx.x;xx.x] | [xx.x;xx.x] |
| Median | XX.X | XX.X | XX.X |
| Q1-Q3 | [xx.x;xx.x] | [xx.x;xx.x] | [xx.x;xx.x] |
| Min-Max | [xx.x;xx.x] | [xx.x;xx.x] | [xx.x;xx.x] |

### 8.6.2.8. Analysis of frequency of access of app pages

A descriptive analysis will be provided by cohort and by intervention arm and overall, on the FAS.

The following template will be used for cohorts 1 and 2 at visits D60, D120 and D180.

| | Cohort 1 |
|--------------------------------------------------------|------------|
| | Enabled |
| | N=XXX |
| The patient use the "report" function | |
| Yes [n (%)] | xx ( xx.x) |
| No [n (%)] | xx ( xx.x) |
| The patient use the "historic of alerts" function | |
| Yes [n (%)] | xx ( xx.x) |
| No [n (%)] | xx (xx.x) |
| The patient use the "log event" function | |
| Yes [n (%)] | xx ( xx.x) |
| No [n (%)] | xx ( xx.x) |
| The patient use his phone to look at his glucose level | |
| Yes [n (%)] | xx ( xx.x) |
| No [n (%)] | xx ( xx.x) |

| Roche Diabetes Care | Statistical Analysis Plan | Dogo 47 / 64 |
|---------------------|---------------------------|---------------------|
| EVERSENSE | Version 2.0 – 30/09/2020 | Page <b>47 / 64</b> |

The following template will be used for cohort 2 at D180 visit.

| | Coh | Cohort 2 | |
|---|---|---|---|
| | Switch | Enabled | Total |
| | N=XXX | N=XXX | N=XXX |
| The patient use the "report" function | | | |
| Yes [n (%)] | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) |
| No [n (%)] | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) |
| The patient use the "historic of | | | |
| alerts" function | | | |
| Yes [n (%)] | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) |
| No [n (%)] | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) |
| The patient use the "log event" | | | |
| function | | | |
| Yes [n (%)] | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) |
| No [n (%)] | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) |
| The patient use his phone to look at | | | |
| his glucose level | | | |
| Yes [n (%)] | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) |
| No [n (%)] | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) |

## 8.6.2.9. Analysis of frequency and type of alarms/alerts received

A descriptive analysis will be provided by cohort and by intervention arm and overall, on the FAS.

The following template will be used.

### Alerts from D0 to D30:

| | Cohort 2 | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | Future Control Future Enabled | | | | | | mo+ol | |
| | Futi | | | Futi | _ | | Total | | |
| | | N=XX | X | | N=XX | X | | N=XX | X |
| | N | | | N | | | N | | |
| | Evt | N | 용 | Evt | N | 용 | Evt | N | 양 |
| READER ALARM | XXX | XX | XX.X | XXX | XX | XX.X | XXX | XX | XX.X |
| Calibration | XXX | XX | XX.X | XXX | XX | XX.X | XXX | XX | XX.X |
| Calibration Expired | XXX | XX | XX.X | XXX | XX | XX.X | XXX | XX | XX.X |
| Calibration Past Due | XXX | XX | XX.X | XXX | XX | XX.X | XXX | XX | XX.X |
| Sensor Glucose | XXX | XX | XX.X | XXX | XX | XX.X | XXX | XX | XX.X |
| Rate Falling | XXX | XX | XX.X | XXX | XX | XX.X | XXX | XX | XX.X |
| Hight Glucose | XXX | XX | XX.X | XXX | XX | XX.X | XXX | XX | XX.X |
| Out of Range High Glucose | XXX | XX | XX.X | XXX | XX | XX.X | XXX | XX | XX.X |
| Out of Range Low Glucose | XXX | XX | XX.X | XXX | XX | XX.X | XXX | XX | XX.X |
| Etc. | XXX | XX | XX.X | XXX | XX | XX.X | XXX | XX | XX.X |
| READER MISC | XXX | XX | XX.X | XXX | XX | XX.X | XXX | XX | XX.X |
| Etc. | | | | | | | | | |

 $\underline{\text{Note}}$ : N Evt = nb of events (i.e. alarms), N = nb of patients with at least one alarm, % = percentage of patients with at least one alarm.

The same template will be used for cohort 1.

| Roche Diabetes Care | Statistical Analysis Plan | Daga 49 / 64 |
|---------------------|---------------------------|---------------------|
| EVERSENSE | Version 2.0 – 30/09/2020 | Page <b>48 / 64</b> |

### Alerts from D30 to D180:

| | Cohort 2 | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | D30-D120 Control | | | D30- | D30-D120 Enabled D30-D180 Enabled | | | | D120-D180 Switch | | | |
| | | N=XXX | ζ | | N=XXX | ζ | | N=XXX | ζ | | N=XXX | ζ |
| | N | | | N | N | | N | | | N | | |
| | Evt | N | 용 | Evt | Evt | N Evt | Evt | N | 용 | Evt | N | 용 |
| READER ALARM | XXX | XX | XX.X | XXX | XXX | XXX | XXX | XX | XX.X | XXX | XX | XX.X |
| Calibration | XXX | XX | XX.X | XXX | XXX | XXX | XXX | XX | XX.X | XXX | XX | XX.X |
| Calibration Expired | XXX | XX | XX.X | XXX | XXX | XXX | XXX | XX | XX.X | XXX | XX | XX.X |
| Calibration Past Due | XXX | XX | XX.X | XXX | XXX | XXX | XXX | XX | XX.X | XXX | XX | XX.X |
| Sensor Glucose | XXX | XX | XX.X | XXX | XXX | XXX | XXX | XX | XX.X | XXX | XX | XX.X |
| Rate Falling | XXX | XX | XX.X | XXX | XXX | XXX | XXX | XX | XX.X | XXX | XX | XX.X |
| Hight Glucose | XXX | XX | XX.X | XXX | XXX | XXX | XXX | XX | XX.X | XXX | XX | XX.X |
| Out of Range High Glucose | XXX | XX | XX.X | XXX | XXX | XXX | XXX | XX | XX.X | XXX | XX | XX.X |
| Out of Range Low Glucose | XXX | XX | XX.X | XXX | XXX | XXX | XXX | XX | XX.X | XXX | XX | XX.X |
| Etc. | XXX | XX | XX.X | XXX | XXX | XXX | XXX | XX | XX.X | XXX | XX | XX.X |
| READER MISC | XXX | XX | XX.X | XXX | XXX | XXX | XXX | XX | XX.X | XXX | XX | XX.X |
| Etc. | | | | | | | | | | | | |

 $\underline{\text{Note}} \colon \text{N Evt} = \text{nb of events (i.e. alarms), N} = \text{nb of patients with at least one alarm, } \% = \text{percentage of patients with at least one alarm.}$ 

The same template will be used for cohort 1 without "D120-D180 Switch" column.

### 8.6.2.10. Analysis of HbA1C (%) level

### HbA1c (%) level at D120 visit:

This endpoint will be analyzed as described for the primary analysis of the cohort 1 primary endpoint, i.e. descriptive analysis and ANCOVA model on the FAS with method 3 (linear interpolation, LOCF and BOCF) for handling of missing data.

The same analysis will be provided for cohort 2.

### HbA1c (%) at D180 visit for cohort 2 only:

This endpoint will be analyzed as described for the primary analysis of the cohort 1 primary endpoint, i.e. descriptive analysis and ANCOVA model on the FAS with method 3 (linear interpolation, LOCF and BOCF) for handling of missing data.

### HbA1c at D120 visit classified as follows: ≤7% / >7%

This endpoint will be analyzed as described for the analysis of % CV < 36% /  $\geq$  36%, section 8.6.2.4.1.

#### HbA1c at D120 visit classified as follows: ≤6.5% / >6.5%

This endpoint will be analyzed as described for the analysis of % CV < 36%,  $\geq$  36%, section 8.6.2.4.1.

#### HbA1c at D180 visit classified as follows: ≤7% / >7%

This endpoint will be analyzed as described for the analysis of % CV < 36%,  $\geq$  36%, section 8.6.2.4.1.

| Roche Diabetes Care | Statistical Analysis Plan | Page <b>49</b> / <b>64</b> |
|---------------------|---------------------------|----------------------------|
| EVERSENSE | Version 2.0 – 30/09/2020 | Page <b>49</b> / <b>64</b> |

### HbA1c at D180 visit classified as follows: ≤6.5% / >6.5%

This endpoint will be analyzed as described for the analysis of % CV < 36% /  $\geq$  36%, section 8.6.2.4.1.

## 8.6.2.11. Maintain of the Eversense effect on hypoglycemia between D150 and D180 for enabled group

This endpoint will be analyzed on patients from the FAS who were randomized in Enabled arm of Cohort 2.

A descriptive analysis will be provided for:

- Percentage of time spent in hypoglycemia <54mg/dL between D90 and D120 visit</li>
- Percentage of time spent in hypoglycemia <54mg/dL between D150 and D180 visit</li>
- Difference in percentage of time spent in hypoglycemia <54mg/dL between (D90-D120) and (D150-D180)

<u>Note:</u> Normality of distribution will be studied using a histogram with the normal probability density curve.

### Main analysis (parametric model):

A restricted maximum likelihood (REML) estimation based on mixed effect model for repeated measures analysis will be used to obtain adjusted means. This model will include time (1="D90-D120", 2="D150-D180") and center as fixed classification effects and the level of hypoglycemia at baseline (percentage of time spent in hypoglycemia <54 mg/dl between D0 visit and D30 visit) as baseline covariates. An unstructured covariance structure will be used to model the within-patient measurements. The Kenward-Roger approximation will be used to estimate denominator degrees of freedom. The comparison of interest will be the contrast between "D90-D120" and "D150-D180". Adjusted means with their 95% CI will be provided. P-values of each effects and covariates will be displayed.

The following template will be used.

| | | Cohort 2 - En | abled arm |
|-----------------------------|-------------|---------------|-------------|
| | Enabled | Enabled | Difference |
| | D90-D120 | D150-D180 | |
| | N=XXX | N=XXX | |
| Percentage of time spent in | | | |
| hypoglycemia <54mg/dL | | | |
| Adjusted mean | XX.X | XX.X | XX.X |
| 95% CI | [xx.x;xx.x] | [xx.x;xx.x] | [xx.x;xx.x] |
| p value | | | p=0.xxx |

From a mixed model for repeated measures including time (1="D90-D120", 2="D150-D180") and Center (p=0.xxx) as fixed classification effect and time spent in hypoglycemia <54 mg/dl between D0 visit and D30 visit (p=0.xxx) as baseline covariate.

### **Sensitivity analysis #1:**

A (non-parametric) Wilcoxon-Mann-Whitney test will be performed.

| Roche Diabetes Care | Statistical Analysis Plan | Dogo <b>FO / 64</b> |
|---------------------|---------------------------|---------------------|
| EVERSENSE | Version 2.0 – 30/09/2020 | Page <b>50 / 64</b> |

### The following template will be used.

| | | Cohort 2 | | |
|---|---|---|---|---|
| | Statistical | Enabled | Enabled | |
| | test | D90-D120 | D150-D180 | Difference |
| | | N=XXX | N=XXX | |
| Percentage of time spent | | | | |
| in hypoglycemia <54mg/dL: | | | | |
| N | | XXX | XXX | XXX |
| Mean (SD) | Wilcoxon | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| Median | p = x.xxx | XX.X | XX.X | XX.X |
| Q1 ; Q3 | | xx.x ; xx.x | xx.x ; xx.x | xx.x ; xx.x |
| Min; Max | | xx.x ; xx.x | xx.x ; xx.x | xx.x ; xx.x |

## 8.6.2.12. Comparison of data from D90-D120 period to D150-D180 period for control group

This endpoint will be analyzed on patients from the FAS who were randomized in Control arm of Cohort 2.

The same analysis as described in section 8.6.2.11 will be provided.

The following template will be used.

| Cohort 2 - Control arm | | |
|---|---|---|
| Control | Switch | Difference |
| D90-D120 | 150-D180 | (control-switch) |
| N=XXX | N=XXX | |
| XX.X | XX.X | xx.x |
| [xx.x;xx.x] | [xx.x;xx.x] | [xx.x;xx.x] |
| | | p=0.xxx |
| | Control D90-D120 N=XXX | Control Switch D90-D120 150-D180 N=XXX N=XXX |

From a mixed model for repeated measures including time (1="D90-D120", 2="D150-D180") and Center (p=0.xxx) as fixed classification effect and time spent in hypoglycemia <54 mg/dl between D0 visit and D30 visit (p=0.xxx) as baseline covariate.

### The following template will be used.

| | | Cohort 2 | | |
|---|---|---|---|---|
| | Statistical | Control | Switch | |
| | test | D90-D120 | D150-D180 | Difference |
| | | N=XXX | N=XXX | |
| Percentage of time spent | | | | |
| in hypoglycemia <54mg/dL: | | | | |
| N | | XXX | XXX | XXX |
| Mean (SD) | Wilcoxon | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| Median | p = x.xxx | XX.X | XX.X | XX.X |
| Q1 ; Q3 | | xx.x ; xx.x | xx.x ; xx.x | xx.x ; xx.x |
| Min; Max | | xx.x ; xx.x | xx.x ; xx.x | xx.x ; xx.x |

### 8.6.2.13. Analysis of Patient Reported Outcome Measures (PROMs)

A descriptive analysis will be provided by cohorts and intervention arm, on the FAS.

Free-text questionnaire will be listed.

| Roche Diabetes Care | Statistical Analysis Plan | Dogo <b>F1</b> / <b>6</b> 4 |
|---|---|---|
| EVERSENSE | Version 2.0 – 30/09/2020 | Page <b>51 / 64</b> |

## 8.6.2.14. Graphical representation of the mean daily glucose level over the 6-month period

The following figure will be provided by cohort.



## 8.7. Safety analysis

All safety analyses will be performed on the Safety Set.

### 8.7.1. Adverse events

### 8.7.1.1. Overall summary of adverse events

An overall summary of TEAEs will be provided by cohort and by intervention arm and overall, for all categories of AE defined in section 6.3.

The following template will be used.

| | Coh | | |
|---|---|---|---|
| | Control<br>N=xxx | Enabled<br>N=xxx | Total<br>N=xxx |
| Patient experiencing at least one AE [n (%)] | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) |
| Patient experiencing at least one TEAE [n (%)] | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) |
| Patient experiencing at least one Serious TEAE [n (%)] | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) |
| TEAE by maximum severity: | | | |
| Mild TEAE | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) |
| Moderate TEAE | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) |
| Severe TEAE | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) |

| | Coh | ort 1 | |
|---|---|---|---|
| | Control<br>N=xxx | Enabled<br>N=xxx | Total<br>N=xxx |
| Detient experiencing at least one Fotal TEAF in (0/ ) | vov ( vov vv) | vv ( vv v) | vov ( vov v) |
| Patient experiencing at least one Fatal TEAE [n (%)] | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) |
| Patient experiencing at least one TEAE leading to discontinuation of the investigational device [n (%)] | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) |
| Patient experiencing at least one TEAE with possible or probable relationship with investigational device [n (%)] | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) |
| Patient experiencing at least one Symptomatic hypoglycemia | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) |
| Patient experiencing at least one Severe hypoglycemia (SAEs) | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) |
| Patient experiencing at least one Serious Diabetic Ketoacidosis (SAEs) | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) |
| Adverse Device Effect (ADE) as collected in eCRF | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) |
| ADEs as reported to the hotline | xx ( xx.x) | xx ( xx.x) | xx ( xx.x) |

This analysis will be done for:

- Cohort 1 from D0 to D180
- Cohort 2 from D0 to D120
- Cohort 2 from D120 to D180
- Cohort 2 from D0 to D180 (for enabled arm only)
- Follow-up arm from D0 to D180.

### 8.7.1.2. Analysis of adverse events by MedDRA coding

A descriptive analysis will be provided by MedDRA SOC and MedDRA PT, by cohort and by intervention arm and overall for the following categories of adverse events:

- AE
- TEAE
- Serious TEAE
- Fatal TEAE
- Related TEAE
- TEAE leading to discontinuation of the investigational device
- Mild TEAE
- Moderate TEAE
- Severe TEAE
- Symptomatic hypoglycemia
- Severe hypoglycemia (SAEs)
- Serious Diabetic Ketoacidosis

Tables will summarize the total number of events and the number and percentage of patients experiencing the event (i.e. in the case of patients experiencing the same event more than once during

| Roche Diabetes Care | Statistical Analysis Plan | Page 53 / 64 |
|---------------------|---------------------------|--------------|

the study, the patient will be counted only once in the same SOC/PT level). The SOC will be sorted by descending frequency and PT will be sorted by descending frequency (within SOC, on « total » column).

| | Cohort 1 | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | _ | ontro | | E<br>( | | | l<br>x) | | |
| System Organ Class / Preferred Term | Nb Nb % Nb Nb %<br>AE pat pat AE pat pat | | | Nb<br>AE | Nb<br>pat | %<br>pat | | | |
| TOTAL | X | X | x.x | X | X | x.x | х | X | x.x |
| SOC A | X | X | x.x | X | x | x.x | х | X | x.x |
| - PT 1 | X | X | x.x | x | X | x.x | x | X | x.x |
| - PT 2 | x | х | x.x | х | х | x.x | x | x | X.X |
| | X | X | x.x | X | X | x.x | X | x | x.x |
| SOC B | X | X | X.X | X | X | x.x | X | X | X.X |
| - PT 1 | X | X | x.x | X | X | x.x | X | X | x.x |
| - PT 2 | x | x | x.x | x | X | x.x | x | x | x.x |
| | X | х | x.x | X | X | x.x | X | X | x.x |

Nb AE = number of adverse events.

Nb pat = number of patients experiencing the event

This analysis will be done for:

- Cohort 1 from D0 to D180
- Cohort 2 from D0 to D120
- Cohort 2 from D120 to D180
- Cohort 2 from D0 to D180 (for enabled arm only)
- Follow-up arm from D0 to D180.

### 8.7.1.3. Analysis of adverse events per 100 patient years

Incidence rates of all AEs and of AEs of special interest (as captured on the AE Form in the eCRF) per 100 patient years will be calculated together with exact two-sided 95% CIs, by cohort and by intervention arm.

This analysis will be done for:

- Cohort 1 from D0 to D180
- Cohort 2 from D0 to D120
- Cohort 2 from D120 to D180
- Cohort 2 from D0 to D180 (for enabled arm only)
- Follow-up arm from D0 to D180.

The following template will be used.

<sup>%</sup> pat = percentage of patients experiencing the event

| Roche Diabetes Care | e Diabetes Care Statistical Analysis Plan | |
|---|---|---|
| EVERSENSE | Version 2.0 – 30/09/2020 | Page <b>54 / 64</b> |

| Cohort 1 | Control | | | | | Enabled | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | N | % | IC 95% | Time at risk<br>(pt-years) | Rate/100 pt-<br>years | N | % | IC 95% | Time at risk<br>(pt-years) | Rate/100<br>pt-years |
| Number of patients | Х | 100 | | | | х | 100 | | | |
| Patient with any AE | Х | XX.X | [xx.x;xx.x] | X.X | xxx.x | х | XX.X | [xx.x;xx.x] | X.X | XXX.X |
| Patient with serious AEs | Х | XX.X | [xx.x;xx.x] | X.X | xxx.x | х | XX.X | [xx.x;xx.x] | X.X | XXX.X |
| Patients with investigator defined investigational related AEs | х | xx.x | [xx.x;xx.x] | X.X | xxx.x | x | xx.x | [xx.x;xx.x] | x.x | xxx.x |
| Patients with AEs leading to discontinuation of investigational device | х | XX.X | [xx.x;xx.x] | X.X | xxx.x | x | XX.X | [xx.x;xx.x] | X.X | XXX.X |
| | | XX.X | | | | | XX.X | | | |
| Adverse Device Effect (ADE) as collected in eCRF | х | xx.x | [xx.x;xx.x] | X.X | xxx.x | х | XX.X | [xx.x;xx.x] | X.X | XXX.X |
| Anticipated ADE as collected in eCRF | х | xx.x | [xx.x;xx.x] | X.X | xxx.x | х | XX.X | [xx.x;xx.x] | X.X | XXX.X |
| Unanticipated ADE as collected in eCRF | х | XX.X | [xx.x;xx.x] | X.X | xxx.x | х | XX.X | [xx.x;xx.x] | X.X | XXX.X |

### Note:

Percentages are calculated using total number of patients per intervention arm as the denominator.

Incidences rates are calculated using number of patients with the respective events per intervention arm divided by time at risk expressed as 100 patient-years.

Patients with AE(s): time at risk = start of first AE – date of first sensor insertion + 1 day.

Patients without AE: time at risk = end of time at risk – date of first sensor insertion + 1 day.

End of time at risk is defined as date of end of studied period (i.e. D120 or D180) or date of premature discontinuation (if it occurs earlier).

| Roche Diabetes Care | Statistical Analysis Plan | Dogo EF / 64 |
|---------------------|---------------------------|--------------|

## 8.8. Individual data listings

All data collected in the CRF will be listed. Individual data listings will be provided in statistical appendices. The following templates will be used.

## 8.8.1. Disposition of patients - all patients

| ID | Sex | Cohort | Date of<br>informed<br>consent | Date of randomization | Date of first<br>sensor insertion | Date of last<br>sensor insertion | Date of completion/<br>Discontinuation | Complet<br>ed<br>study? | Reason for<br>not<br>performing<br>following-<br>up | Extent of exposure (days) |
|---|---|---|---|---|---|---|---|---|---|---|
| СххРххх | М | 1 | yyyy-mm-dd | уууу-mm-dd | уууу-mm-dd | yyyy-mm-dd | yyyy-mm-dd | Yes | | xxx |
| СжжРжжж | F | 2 | уууу-mm-dd | уууу-mm-dd | уууу-mm-dd | yyyy-mm-dd | yyyy-mm-dd | No | Lost to<br>follow-up | ххх |
| | | | | | Number o | f patients = xxx | | | | |

## 8.8.2. Protocol deviations - all patients

| I | ID | | IN/EX criteria not respected or missing | |
|---|---|---|---|---|
| Center | Center Patient Criterion number | | | |
| | | IN 2 Male and female patients at least 18 years of age | | No |
| | ЕХ 3 | | History of hepatitis B, hepatitis C, or HIV | Yes |
| | (. | | () | () |
| | | () | () | () |
| () | ) () () | | () | () |

| Roche Diabetes Care | Statistical Analysis Plan | Page 56 / 64 |
|---------------------|---------------------------|--------------|

### 8.8.3. Analysis sets and cohorts analyzed - all patients

| I | D | | Analysis sets | | | | |
|---|---|---|---|---|---|---|---|
| Center | Center Patient | | Screened Set | Randomized Set | Safety Set | Full Analysis set | Per Protocol |
| | | 1 | Yes | Yes | Yes | Yes | Yes |
| | | 2 | Yes | Yes | No | No | No |
| () | () | | | | | | |
| () | () | | | | | | |

### 8.8.4. Demographic data and other baseline characteristics, including medical history and therapies – all patients

| Center-Patient | Sex | Diabetes type | Of childbearing capacity | Urine pregnancy<br>test done | Result | Date of birth | Weight (kg) | Height (cm) | BMI (kg/m²) |
|---|---|---|---|---|---|---|---|---|---|
| СжжРжжж | Male | 1 | Y | Y | Negative | ттуууу | xxx | xxx | ххх |
| CxxPxxx | Female | 2 | N | | | ттуууу | xxx | xxx | xxx |

The same template as above will be used for:

- Diabetes history (i.e. diabetes duration, type of diabetes, usual self-monitoring blood glucose: capillary blood glucose monitoring or flash glucose monitoring, etc.)
- Diabetes complications
- Last HbA1c analysis
- Diabetes Family History
- Diabetes Medication
- Medical history diseases other than Diabetes
- Previous medications for diseases other than Diabetes
- Training at sensor insertion (D0) (arm chosen for insertion, trainer, etc.)
- Training to the device after randomization (at D30) for Enabled group

| Roche Diabetes Care | Statistical Analysis Plan | Dogo 57 / 64 |
|---------------------|---------------------------|--------------|

- Age (years)
- BMI
- Time since start of diabetes (years)
- Time since last blood test for HbA1c (days)
- Duration of insertion procedure (minutes)
- Duration of removal procedure (minutes)

## 8.8.5. Extent of exposure and treatment compliance

Individual data listings will be provided on the SAF.

## 8.8.6. Primary efficacy endpoint

## 8.8.6.1. Cohort 1: HbA1c (%) level - RS

| ID | Cohort | FAS | PP | SAF | HbAlc (%) level | | |
|---------|--------|-----|----|-----|-----------------|------|------|
| | | | | | D0 | D120 | D180 |
| CxxPxxx | 1 | Y | Y | Y | xx | xx | xx |
| СжжРжжж | 1 | Y | Y | Y | xx | xx | xx |
| Etc. | Etc. | | : | : | | | |

## 8.8.6.2. Cohort 2: percentage of time in hypoglycemia <54mg/dL between D90 visit and D120 visit - RS

| ID | Cohort | RS | FAS | PP | SAF | Time (%) between D90 and D120 | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | <54 mg/dL | <70 mg/dL | Euglycemia | >180 mg/dL | >250 mg/dL |
| CxxPxxx | 2 | Y | Y | Y | Y | xx | xx | xx | xx | xx |
| CxxPxxx | 2 | Y | Y | Y | Y | xx | xx | xx | xx | xx |
| Etc. | Etc. | | | | | | | | | |

| Roche Diabetes Care | Statistical Analysis Plan | Page <b>58 / 64</b> |
|---------------------|---------------------------|---------------------|

## 8.8.7. Secondary efficacy endpoint

The same template as above will be used for all secondary efficacy endpoints.

### 8.8.8. Adverse events

All AEs will be listed on the RS.

| Roche Diabetes Care | Statistical Analysis Plan | Do 20 FO / CA |
|---------------------|---------------------------|---------------------|
| EVERSENSE | Version 2.0 – 30/09/2020 | Page <b>59 / 64</b> |

### 9. **ALGORITHMS**

### 9.1. Handling of missing CGM data

Fig. 1 is designed to understand how the algorithm operates for the replacement of missing CGM data.



Figure 1. Daily Glucose

### **Case 1:**

Glycemia values below 40 mg/dL are marked as "Out of Physiological Range" in the CGM files and recorded as missing values. In addition, the first record below 40 mg/dL is marked as "Out of Range Low Glucose". The following records are only marked as "Out of Physiological Range" without further details, until glycemia values returns within detection range.

These missing data will be replaced as described below:

- Missing data flagged as "Out of Range Low Glucose" by CGM system will be imputed to 40 mg/dL
- 2. Missing data flagged as "Out of Physiological Range" by CGM system will be imputed to <u>40</u> <u>mg/dL</u> under the following conditions:
  - a. If the "Out of Physiological Range" missing data is within 30 minutes <u>after</u> an available value that is smaller than 70 mg/dL,
  - b. If the "Out of Physiological Range" missing data is within 30 minutes **before** an available value that is smaller than 70 mg/dL,
  - c. If the "Out of Physiological Range" missing data is within 30 minutes <u>after</u> an "Out of Physiological Range" value already imputed to 40 mg/dL,
  - d. If the "Out of Physiological Range" missing data is within 30 minutes **before** an "Out of Physiological Range" value already imputed to 40 mg/dL.

| Roche Diabetes Care | Statistical Analysis Plan | Dogo 60 / 64 |
|---------------------|---------------------------|---------------------|
| EVERSENSE | Version 2.0 – 30/09/2020 | Page <b>60 / 64</b> |

#### Case 2:

Glycemia values above 400 mg/dL are marked as "Out of Physiological Range" in the CGM files and recorded as missing values. In addition, the first record above 400 mg/dL is marked as "Out of Range High Glucose". The following records are only marked as "Out of Physiological Range" without further details, until glycemia values returns within detection range.

These missing data will be replaced as described below:

- Missing data flagged as "Out of Range High Glucose" by CGM system will be imputed to 400 mg/dL
- 2. Missing data flagged as "Out of Physiological Range" by CGM system will be imputed to <u>400</u> mg/dL under the following conditions:
  - a. If the "Out of Physiological Range" missing data is within 30 minutes <u>after</u> an available value that is greater than 180 mg/dL,
  - b. If the "Out of Physiological Range" missing data is within 30 minutes **before** an available value that is greater than 180 mg/dL,
  - c. If the "Out of Physiological Range" missing data is within 30 minutes <u>after</u> an "Out of Physiological Range" value already imputed to 400 mg/dL,
  - d. If the "Out of Physiological Range" missing data is within 30 minutes **before** an "Out of Physiological Range" value already imputed to 400 mg/dL.

Note: an "Out of Physiological Range" data that can be imputed both to 40 mg/dL according to rule 1 and 400 mg/dL according to rule 2 will not be replaced.

### Cases 3 and 4:

It is expected that glycemia values are recorded every 5 minutes by CGM system. However, there can be more than 5 minutes between 2 consecutive records (e.g. temporary discontinuation, discharged battery, transmitter temporarily removed, etc.). A threshold of 30 minutes between 2 consecutive records has been defined. CGM data will be handled as described below whether there is more or less than 30 minutes between 2 consecutive records:

- 1. If 30 minutes or more between 2 consecutive records: this is considered as a temporary discontinuation of the CGM system (no interpolation nor any other approach of replacement).
- 2. If less than 30 minutes between 2 consecutive records: linear interpolation will be used for calculation of time spent (cf. next section).

# 9.2. Computation rules for time spent in-, below- and above- target ranges

The algorithm can be adjusted to:

- Targeted range of glucose values: lower and upper limit,
- Specified time interval: start time and end time for analysis.
- Maximum allowed duration (min) between 2 records (30 min by default)

After replacement of missing data flagged as "Out of Physiological Range", the algorithm will automatically compute time in-, below- or above- the targeted range of glucose values for the given duration.

| Roche Diabetes Care | Statistical Analysis Plan | Dogo 61 / 64 |
|---------------------|---------------------------|----------------------------|
| EVERSENSE | Version 2.0 – 30/09/2020 | Page <b>61</b> / <b>64</b> |

**Example 1:** Referring to figure 2, for the period between the start point and the end point, the algorithm gives the following results:

• Hyperglycemia: 0.5 + 2 = 2.5 hours

• Euglycemia: 4 + 2 = 6 hours

• Hypoglycemia: 2 hours

Non-replaced missing data: 2 hours



Figure 2. Pattern for computation rules

### Example 2:

Assuming we have the following data for a patient after running the algorithm and for a period of 24h:

Hyperglycemia: 4 hoursEuglycemia: 14 hoursHypoglycemia: 2 hours

- Non-replaced missing data: 4 hours

Computation of time spent in range values gives the percentage of time in:

Hyperglycemia: (4/20)\*100 = 20%
 Euglycemia: (14/20)\*100 = 70%
 Hypoglycemia: (2/20)\*100 = 10%.

Availability of sensor data: (20/24)\*100 = 83%.

| Roche Diabetes Care | Statistical Analysis Plan | Daga 62 / 64 |
|---------------------|---------------------------|----------------------------|
| EVERSENSE | Version 2.0 – 30/09/2020 | Page <b>62</b> / <b>64</b> |

# 10. CHANGES IN THE STATISTICAL METHODS FROM THOSE STATED IN THE PROTOCOL

This Statistical Analysis Plan is based on Protocol V5.0 dated of 11/12/2018 and CRF V2.0.1 dated 24/04/2019.

### Clarification about Section 14.4 of the Protocol:

It is stated in the Protocol, Section 14.4 (Analysis of the primary endpoint for cohort 2): "In case of non-normal distribution, a study will be done in order to use either a model based on **Poisson distribution** or a non-parametric test approach".

Since the primary endpoint of cohort 2 is a continuous data, Poisson distribution is not appropriate (Poisson is appropriate for count data only).

Therefore, this sentence has been interpreted in the SAP as follows: "In case of non-normal distribution, a study will be done in order to use either a model based on **non-normal parametric distribution** or a non-parametric test approach".

### Analysis planned in the Protocol not performed:

It is stated in the Protocol, Section 14.6 (Safety analysis): "The following ADEs are of particular interest: ADEs and unanticipated ADEs leading to replacement of device. Incidence rates of all ADEs and of these ADEs and AEs of special interest (as captured on the AE Form in the eCRF) per 100 patient years will be calculated together with exact two-sided 95% CIs assuming that the number of special AEs observed in the study is Poisson distributed".

ADEs leading to replacement of device will not be analyzed, as it was not collected in the eCRF whether ADE led to replacement of device or not.

There are no other changes in the statistical methods from those stated in the protocol.

| Roche Diabetes Care | Statistical Analysis Plan | Dogo 62 / 64 |
|---------------------|---------------------------|---------------------|
| EVERSENSE | Version 2.0 – 30/09/2020 | Page <b>63 / 64</b> |

## 11. QUALITY CONTROL

A self-validation will be performed by the statistician in charge of the analysis as follows: each derived variables will be validated exhaustively (i.e. on all patients) whenever possible. Exhaustive controls can be performed using either contingency tables (i.e. displaying all qualitative variables and minimum/maximum values of quantitative variables involved in the derivation rules) or individual data listings that are considered as not too large (i.e. no more than 50 rows). An exhaustive control is considered possible when the corresponding output contains up to 50 rows. For validation outputs considered as too large (i.e. more than 50 rows), the validation can be performed on a minimum of 5% patients randomly drawn. If the validation output is still too large (i.e. more than 50 rows), the validation will be performed on a subset of 50 rows (minimum).

Validation outputs will be review by a third party (i.e. head of biostatistics or another statistician).

In particular, derivation of the primary endpoint will be double-checked by a third party (i.e. head of biostatistics or another statistician).

| Roche Diabetes Care | Statistical Analysis Plan | Dogo 64 / 64 |
|---------------------|---------------------------|---------------------|
| EVERSENSE | Version 2.0 – 30/09/2020 | Page <b>64 / 64</b> |

## 12. References

- 1. Toward Defining the Threshold Between Low and High Glucose Variability in Diabetes. Louis Monnier, Claude Colette, Anne Wojtusciszyn, Sylvie Dejager, Eric Renard, Nicolas Molinari, David R. Owens. 7, Diabetes Care Jul 2017, Vol. 40, pp. 832-838.
- 2. Are risk indices derived from CGM interchangeable with SMBG-based indices? **Fabris C, Patek SD, Breton MD.** 2015, J Diabetes Sci Technol., pp. 50-59.